Humira® for subcutaneous use only

Special drug-use survey

-Long-term survey on Colitis ulcerative-

Statistical Analysis Plan (the 6th periodical safety report/re-examination/final report)

Version 2.1

Prepared in 2018 March 12

1. Approval

Entruster

Company name AbbVie GK

Approved by Post-marketing Surveillance Supervisor Seal

Date of approval MMM, DD, YYYY

Approved by Medical Supervisor Seal

Date of approval MMM, DD, YYYY

Approved by Safety Management Supervisor Seal

Date of approval MMM, DD, YYYY

Approved by Survey Planning Physician Seal

Date of approval MMM, DD, YYYY

Approved by Statistical Analysis Supervisor Seal

Date of approval MMM, DD, YYYY

Entruster

Company name Eisai Co., Ltd.

Approved by Neurology Medical Department, Statistical Analysis Supervisor Seal

Date of approval MMM, DD, YYYY

Entrustee

Company name A2 Healthcare Corporation

Approved by Statistical Analysis Project Leader Seal

Date of approval MMM, DD, YYYY

### Table of Contents

| 1. I | Preparation/revision history | 10 |
|---|---|---|
| 2. I | Definitions of terms and abbreviations | 16 |
| 3. ( | Objective of this statistical analysis plan | 17 |
| 3.1 | . Objective of developing this statistical analysis plan | 17 |
| 4. 7 | The survey outline | 17 |
| 4.1 | . Survey objective | 17 |
| 4.2 | . Survey plan | 17 |
| 4.3 | . Target sample size for the survey | 17 |
| 5. I | tems to be analyzed and the methods | 19 |
| 5.1 | . Analysis items | 19 |
| 5.2 | . Analysis method | 20 |
| 6. I | Presence/absence of analysis and its schedule | 20 |
| 7. S | Softwares/dictionary used for analysis | 21 |
| 7.1 | . Statistical analysis and listing softwares | 21 |
| 7.2 | . Dictionary for use | 21 |
| 8. | The definition of the groups used for analysis | 22 |
| 9. ( | General agreement items for analysis | 23 |
| 9.1 | . Handling of missing data | 23 |
| 9.2 | . Descriptive statistics | 23 |
| 9.3 | . Display digit for figures | 24 |
| 9.4 | . Figure display rule | 24 |
| 9.5 | . Statistical test method | 24 |
| 9.6 | . Significant level | 24 |
| 10. I | Derivation and calculation methods for data | 25 |
| 10. | 1. General | 25 |
| 1 | Number of site | 25 |
| 1 | Number of patients per site | 25 |
| F | Patients with an adverse event which occurred not in the safety analysis period | 25 |
| | Patients who developed an infection | |
| F | Patients who developed tuberculosis | 25 |
| F | Patients who developed malignant tumour | 25 |
| F | Patients who developed an administration site reaction | 25 |
| F | Patients who developed an autoimmune disease | 25 |
| F | Patients who developed pancytopenia | 25 |
| F | Patients who developed demyelinating disease | 25 |
| | Patients who developed cardiac failure congestive | |
| F | Patients who developed interstitial pneumonia | 25 |

| Patients subject to AAA measurement | 25 |
|----------------------------------------------------------------------|----|
| Patients of contraindications | 26 |
| The first administration date of Humira. | 26 |
| The final administration date of Humira | 26 |
| Days to the final administration date of Humira | 27 |
| Administration status (dosage and administration) | 27 |
| Reason for change in dose/dosing frequency | 28 |
| Administration status (total number of dosing, total dose) | 28 |
| Discontinued patients | 29 |
| Presence/absence of reason for discontinuation | 29 |
| Reason for discontinuation | 29 |
| Reason for discontinuation, other reasons | 29 |
| Patients who continue the survey | 29 |
| Presence/absence of complications | 30 |
| Presence/absence of medical history | 30 |
| Complication/Hepatic function disorder | 30 |
| Complication/Renal impairment | 30 |
| Presence/absence of Complication/Circulatory disorder | 30 |
| Presence/absence of Complication/Blood disorder | 30 |
| Presence/absence of Complication/Respiratory disorder | 30 |
| Presence/absence of Complication/others | 30 |
| Medical history: presence/absence of tuberculosis | 31 |
| Medical history: presence/absence of non-tuberculous mycobacteriosis | 31 |
| Medical history: presence/absence of interstitial pneumonia | 31 |
| Medical history: presence/absence of bronchitis bacterial | 31 |
| Medical history: presence/absence of aplastic anaemia | 31 |
| Medical history: presence/absence of pancytopenia | 31 |
| Medical history: presence/absence of malignant tumour | 31 |
| Medical history: presence/absence of other medical history | 31 |
| Presence/absence of allergy history | 32 |
| Patients with an hepatitis B virus infection | 32 |
| Presence/absence of smoking history | 32 |
| Detailed classification of smoking history | 32 |
| Patients with dosing deviation of Humira. | 32 |
| Presence/absence of self-administration | 32 |
| Presence/absence of self-administration error | 33 |
| Sex | 33 |
| Pregnancy/nursing | 33 |

| Race | 33 |
|-----------------------------------------------------------------------|----|
| Age | 33 |
| Pediatrics | 33 |
| The elderly | 33 |
| Body weight | 34 |
| Body height | 34 |
| BMI | 34 |
| Duration of illness (in years) | 34 |
| Indication | 34 |
| Site of disease | 34 |
| HBs antigen test | 34 |
| HBs antibody test | 34 |
| HBc antibody test | 34 |
| HBV-DNA quantification assay | 35 |
| Tuberculin test or IGRA | 35 |
| Chest X ray test | 35 |
| Chest CT test | 35 |
| Other imaging | 35 |
| Chest X ray or CT test | 35 |
| Presence/absence of prior medications | 35 |
| Presence/absence of prior medication (aminosalicylic acid drug) | 36 |
| Presence/absence of prior medication (corticosteroids) | 36 |
| Presence/absence of prior medication (azathioprine) | 36 |
| Presence/absence of prior medication (6-mercaptopurine) | 36 |
| Presence/absence of prior medication (azathioprin & 6-mercaptopurine) | 36 |
| Presence/absence of prior medication (tacrolimus & ciclosporin) | 36 |
| Presence/absence of prior medication (antibiotics) | 36 |
| Presence/absence of prior medication (others) | 37 |
| Presence/absence of prior medication (Infliximab) | 37 |
| Presence/absence of prior medication (other biological products) | 37 |
| Presence/absence of treatment history with biological products | 37 |
| Presence/absence of prior treatment | 37 |
| Presence/absence of prior treatment (surgery) | 37 |
| Presence/absence of prior treatment (leukocytapheresis) | 38 |
| Presence/absence of prior treatment (enteral nutrition therapy) | |
| Presence/absence of prior treatment (intravenous nutrition therapy) | |
| Presence/absence of prior treatment (other therapy) | |
| Presence/absence of concomitant medication | |

| Presence/absence of concomitant medication (aminosalicylic acid drug) | 40 |
|---|---|
| Presence/absence of concomitant medication (corticosteroids) | 40 |
| Presence/absence of concomitant medication (azathioprine) | 40 |
| Presence/absence of concomitant medication (6-mercaptopurine) | 41 |
| Presence/absence of concomitant medication (azathioprine & 6-mercaptopurine) | 41 |
| Presence/absence of concomitant medication (tacrolimus & ciclosporin) | 41 |
| Presence/absence of concomitant medication (antibiotics) | 41 |
| Presence/absence of concomitant medication (others) | 41 |
| Presence/absence of administration of anti-hepatitis B virus agent | 41 |
| Presence/absence of concomitant therapy | 41 |
| Presence/absence of concomitant therapy (surgery) | 42 |
| Presence/absence of concomitant therapy (leukocytapheresis) | 42 |
| Presence/absence of concomitant therapy (enteral nutrition therapy) | 42 |
| Presence/absence of concomitant therapy (intravenous nutrition therapy) | 42 |
| Presence/absence of concomitant therapy (other therapy) | 42 |
| Tuberculosis test | 43 |
| Hepatitis B test | 43 |
| 10.2. Safety analysis | 43 |
| Adverse event | 43 |
| Seriousness of adverse events | 43 |
| Adverse reaction | 43 |
| Serious adverse reactions | 44 |
| Outcome | 44 |
| Death case | 44 |
| Days from the first administration date of Humira to the adverse-event onset date. | 44 |
| Days from the adverse-event onset date to the outcome confirmation date | (recovered or |
| recovering) | 44 |
| Incidence of adverse reactions, incidence of serious adverse reactions, inciden | ce of adverse |
| events, incidence of serious adverse events | 45 |
| 10.3. Effectiveness analysis | 45 |
| General improvement rate | 45 |
| Mayo score | 45 |
| Remission of Mayo score | 45 |
| Partial Mayo score | 45 |
| Remission of partial Mayo score | 45 |
| Improvement of partial Mayo score (responder) | 45 |
| Endoscopy results | 45 |
| 1 How to stratify data | 46 |

| 12. Hand | dling of data for test/assessment periods | 49 |
|---|---|---|
| 12.1. | Assessment period for the administration status of Humira | 49 |
| 12.2. | Assessment period for the onset status of adverse reactions | |
| 12.3. | Assessment period for Mayo score | 50 |
| 12.4. | Assessment period for partial Mayo score | 50 |
| 12.5. | Assessment period for general improvement rate | 50 |
| 12.6. | Assessment period for CRP | 51 |
| 12.7. | Assessment period for the continued administration of Humira | 51 |
| 13. Char | ts to be generated (chart No., chart name) | 52 |
| 13.1. | General | 52 |
| "1.1 | Case structure chart' | 52 |
| "1.2 | The number of sites for survey and the number of patients surveyed" | 52 |
| "1.3 | A list of the patients excluded from the safety analysis group and the patient | s excluded |
| from | the effectiveness analysis group (including the reason for exclusion)" | 52 |
| "1.3. | 1. Excluded patients (aggregation by reason) | 52 |
| "1.4 | A list of patients (adverse event + search flag)" | 53 |
| "1.4. | 1 A list of adverse events" | 54 |
| "1.4. | 2 A list of death cases" | 54 |
| "1.4. | 3 A list of prior/concomitant medications in patients with an CMV infection" | 54 |
| "1.4. | 4 A list of patients aged 18 years or younger" | 54 |
| "1.5 | Administration status of Humira (dosage and administration)" | 55 |
| "1.5. | 1 other dosage and administration (a list)" | 55 |
| "1.6 | Administration status of Humira (dosing frequency, dose) | 55 |
| "1.6. | 1 Administration status of Humira (period)" | 56 |
| "1.6. | 2 Continuation rate of Humira" | 56 |
| "1.7 | Administration status of Humira (discontinuation of administration)" | 56 |
| "1.7. | 1 Administration status of Humira (reason for discontinuation other reasons) | 57 |
| "1.12 | 2 Distribution status of patient backgrounds" | 57 |
| "1.13 | 3 Incidence of self-administration error" | 58 |
| "1.16 | 6 A list of patients with AAA measured | 58 |
| 13.2. | Safety | 58 |
| "2.1 | A list of onset status of adverse reactions/infections (Attachment Form 2) " | 58 |
| "2.1. | 1 A list of the onset status of adverse reactions/infections (patients not in | the safety |
| analy | ysis)" | 59 |
| "2.1. | 2 A list of the onset status of adverse reactions/infections not in the follow-up pe | riod"59 |
| "2.2 | A list of the onset status of serious adverse events (Attachment Form 10)" | 59 |
| "2.3 | A list of target-patient summary (Attachment Form 3)" | 60 |
| "2.4. | 1 A list of the onset status of adverse reactions (priority survey items)" | 62 |

| "2.4.2 A list of the onset status of adverse reactions (identified important risks)"63 |
|---|
| "2.4.3 A list of the onset status of adverse events (priority survey items)"64 |
| "2.4.4 A list of the onset status of adverse events (identified important risks)"64 |
| "2.5 A list of the onset status of adverse reactions with/without self-administration"64 |
| "2.5.1 A list of the onset status of adverse reactions with/without self-administration"64 |
| "2.6 Incidence of adverse reactions per onset period (serious)"65 |
| "2.7 Incidence of adverse reactions per set period" |
| "2.9 Incidence of adverse reactions (serious adverse reactions/adverse reactions) per |
| background factor" |
| "2.9.xx Incidence of adverse reactions per background factor and seriousness"66 |
| "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness" |
| "2.14.1 Incidence of adverse reactions with/without renal impairment and per seriousness"67 |
| "2.15.1 Incidence of adverse reactions per seriousness in pediatrics and non-pediatrics"67 |
| "2.16.1 Incidence of adverse reactions per seriousness in the elderly and non-elderly patients" |
| 68 |
| "2.17 A list of the onset status of adverse reactions/infections in this survey" |
| "2.18 A list of the onset status of adverse reactions with/without treatment history with |
| biological products" |
| "2.18.1 A list of the onset status with/without treatment history with biological products |
| (patients excluded from the safety analysis group)"69 |
| "2.19 A list of the onset status of adverse events in this survey" |
| "2.20 A list of the onset status of adverse reactions (all cases)" |
| 13.3. Effectiveness |
| "3.1.1 Changes in Mayo score (Observed Case)" |
| "3.1.2 Changes in the remission rate at each point of Mayo score (Observed Case)"70 |
| "3.1.4 Changes in partial Mayo score (Observed Case)" |
| "3.1.5.1 Changes in the remission rate at each point of partial Mayo Score (Observed Case)".71 |
| "3.1.5.2 Changes in the remission rate (NRI) at each point of partial Mayo Score"72 |
| "3.1.7.1 Remission rate at Week 52 in patients who achieved a remission at Week 8 of |
| administration based on partial Mayo score" |
| "3.1.7.2 Remission rate at Week 52 in patients who achieved the response as an index of partial |
| Mayo score at Week 8 of administration" |
| "3.2 General improvement rate" |
| "3.4 Aggregation for effectiveness per patient background factor (general improvement rate)"73 |
| "3.4.1 Aggregation for effectiveness per patient background factor (partial Mayo score)"74 "3.5 Changes in CPR level" |
| "3.6 The status of corticosteroid use and the remission in partial Mayo score in patients who |

| used corticosteroids when administration was s | tarted (Observed Case)"75 |
|------------------------------------------------|---------------------------|
| "3.7 Endoscopy results during administration p | eriod"75 |

# 1. Preparation/revision history

| Version | Date of | Prepared/revised | D. |
|---|---|---|---|
| No. | preparation/revision | by | Reasons |
| 1.0 | February 6, 2017 | Yutaro Shiraishi | First version |
| 1.1 | May 23, 2017 | Yutaro Shiraishi | ■ General |
| | | | Names of external files were amended |
| | | | for re-examination |
| | | | ■ 2. Definitions of terms and |
| | | | abbreviations |
| | | | • The definitions of "adverse events in |
| | | | the safety analysis period" and "adverse |
| | | | events not in the safety analysis period" |
| | | | were changed |
| | | | ■ 6. Presence/absence of analysis and its |
| | | | schedule |
| | | | • the 7th periodical safety report was |
| | | | deleted. |
| | | | ■ 8. Definitions of groups used for |
| | | | analysis |
| | | | • The definition of "registered patients" |
| | | | was changed, and the definitions of |
| | | | "patients ineligible for registration", |
| | | | "patients with registration pending" and |
| | | | "patients eligible for registration" were |
| | | | deleted. |
| | | | • The definitions of "patients whose |
| | | | survey form was locked" and "patients |
| | | | whose survey form was yet to be locked" |
| | | | were changed. |
| | | | The definition of "patients excluded |
| | | | from the effective analysis group" was |
| | | | partly deleted. |
| | | | ■ 10.1 General |
| | | | • The definition of "reasons for change |
| | | | in dose/dosing frequency" was changed. |
| | | | • Descriptions of "presence of |

| Version | Date of | Prepared/revised | Dangang |
|---|---|---|---|
| No. | preparation/revision | by | Reasons |
| | | | complications", "presence of medical |
| | | | history", "presence of |
| | | | complication/others" and "presence of |
| | | | medical history/others" were amended for |
| | | | clarification |
| | | | • The definitions of "HBs antigen test", |
| | | | "HBs antibody test", "HBc antibody test", |
| | | | "HBV-DNA quantification test" and |
| | | | "Tuberculin test or IGRA test" were |
| | | | changed |
| | | | • The definitions of "Chest X ray or CT |
| | | | test", "tuberculosis test" and "Hepatitis B |
| | | | test" were added |
| | | | • "To describe the drug name" was |
| | | | added to the definitions of "presence of |
| | | | prior medication" and "presence of |
| | | | concomitant medication" |
| | | | ■ 11. How to stratify data |
| | | | • "Circulatory disorders" was deleted in |
| | | | "Detailed classification of complications" |
| | | | "Gastrointestinal disorder" and |
| | | | "Collagen disorder" were deleted in |
| | | | "Other classifications of complications" |
| | | | • "Presence of decreased response", |
| | | | "acute events", "delayed events" and |
| | | | "Unknown/Not provided" were deleted in |
| | | | "Detailed classification of 'using' |
| | | | biological products" |
| | | | ■ 13.1 General |
| | | | • Analysis items of 1.1, 1.3.1, 1.4 and |
| | | | 1.4.1 were changed |
| | | | • 1.4.4 was added |
| | | | • Analysis target in 1.7 and 1.13 was |
| | | | changed |
| | | | Analysis target and items were |

| Version | Date of | Prepared/revised | |
|---|---|---|---|
| No. | preparation/revision | by | Reasons |
| | | - | changed in 1.12. |
| | | | • Analysis target in 3.6 was changed |
| | | | and the table number was also changed to |
| | | | 1.6.2 |
| | | | ■ 13.2 Safety |
| | | | • Analysis items of 2.4.1, 2.4.2, 2.4.3, |
| | | | 2.4.4, 2.9 and 3.4 were changed |
| | | | • 2.5.1, 2.9.xx, 2.18.1 and 2.19 were |
| | | | added. |
| | | | • Remarks were added in 2.6 |
| | | | Analysis target, analysis objective and |
| | | | analysis items were changed in 3.4.1. |
| 2.0 | February 6, 2018 | Yutaro Shiraishi | ■ General |
| | | | Names of external files were amended |
| | | | for final report |
| | | | ■ 6. Presence/absence of analysis and its |
| | | | schedule |
| | | | Final report period was added |
| | | | ■ 7.2. Dictionary in use |
| | | | MedDRA/J version update |
| | | | ■ 8. Definitions of groups used for |
| | | | analysis |
| | | | • Exclusion items for "patients excluded |
| | | | from the efficacy analysis group" were |
| | | | added. |
| | | | ■ 9.3. Digits displayed for figures |
| | | | Descriptions on CRP were added |
| | | | ■ 10.1 General |
| | | | • The definition of "Administration |
| | | | status (dosage and administration)" was |
| | | | amended. |
| | | | • "Reasons for discontinuation/other |
| | | | reasons", "detailed classification of |
| | | | smoking history", "presence of prior |
| | | | medication (azathioprine & |

| Version | Date of | Prepared/revised | Reasons |
|---|---|---|---|
| No. | preparation/revision | by | Reasons |
| | | | 6-mercaptopurine)", "presence of prior |
| | | | medication (tacrolimus & ciclosporin)", |
| | | | "presence of combination drug |
| | | | (azathioprine & 6-mercaptopurine)", and |
| | | | "presence of combination drug (tacrolimus |
| | | | & ciclosporin)" were newly added. |
| | | | • The description of "presence of |
| | | | smoking history" was amended for |
| | | | clarification. |
| | | | The conditions for drug code were |
| | | | added in "presence of prior medication" |
| | | | and "presence of presence of concomitant |
| | | | medication" |
| | | | • "Presence of prior medication |
| | | | (aminosalicylic acid drug)", "presence of |
| | | | prior medication (corticosteroids)", |
| | | | "presence of prior medication |
| | | | (azathioprine)", "presence of prior |
| | | | medication (6-mercaptopurine)", and |
| | | | "presence of prior medication |
| | | | (antibiotics)", were added for the |
| | | | conditions of the survey form. |
| | | | The condition of ciclosporin was |
| | | | added in "presence of prior medication |
| | | | (others)" and "concomitant medication |
| | | | (others)". |
| | | | ■ 10.3 Effectiveness analysis |
| | | | • "Responder of partial Mayo score" |
| | | | was newly added |
| | | | Endoscopy results were added |
| | | | ■ 11. How to stratify data |
| | | | • "Reasons for discontinuation/other |
| | | | reasons", "detailed classification of |
| | | | smoking history" and "disease site per |
| | | | type" were newly added. |

| Version | Date of | Prepared/revised | Reasons |
|---|---|---|---|
| No. | preparation/revision | by | Reasons |
| | | | Azathioprine & 6-mercaptopurine |
| | | | were added and tacrolimus was replaced |
| | | | with tacrolimus & ciclosporin in "detailed |
| | | | classification of prior medications for |
| | | | colitis ulcerative" and "detailed |
| | | | classification of concomitant medications |
| | | | for colitis ulcerative" |
| | | | • "Unknown/Not provided" was added |
| | | | in the discontinuation reason for the |
| | | | detailed classification of 'using' biological |
| | | | products". |
| | | | • "Normal or remission-phase mucosa, |
| | | | mild, moderate, severe in severity" was |
| | | | added in "endoscopy results" |
| | | | ■ 12.3 Assessment period of Mayo score |
| | | | • The definitions of the time of |
| | | | discontinuation and the time of final |
| | | | assessment were added. |
| | | | ■ 12.4 Assessment period of partial Mayo |
| | | | score |
| | | | Time point was added |
| | | | ■ 12.6 Assessment period of CRP |
| | | | Time point was added |
| | | | ■ 12.7 Assessment period for the |
| | | | continued administration of Humira |
| | | | Time point was added |
| | | | ■ 13.1 General |
| | | | • Analysis items of 1.4, 1.4.1, 1.4.4 and |
| | | | 1.12 were changed |
| | | | • Analysis target was changed in 1.6.2 |
| | | | Aggregation details was changed in |
| | | | 1.7.1 |
| | | | ■ 13.2 Safety |
| | | | • The period classification was changed |
| | | | in 2.1 |

| Version No. | Date of preparation/revision | Prepared/revised by | Reasons |
|---|---|---|---|
| | proparation to vision | | <ul> <li>Analysis items were changed in 2.9 and 2.20</li> <li>13.3 Effectiveness</li> <li>3.1.5.2, 3.1.7.2, 3.6 and 3.7 were newly added</li> <li>Analysis details was changed in 3.1.7.1 and 3.4</li> <li>Analysis objective was changed in 3.5</li> <li>Analysis item was changed in 3.5</li> <li>Analysis target and objective were changed in 3.4.1</li> </ul> |
| 2.1 | March 12, 2018. | Yutaro Shiraishi | ■ 11. How to stratify data • "Partial Mayo score" was changed Changed from "≥6 and <9" to "≥6 and ≤9" |

# 2. Definitions of terms and abbreviations

The terms and abbreviations used in this analysis plan are as follows:

| Term and abbreviation | Definition |
|---|---|
| | Any untoward or unintended symptoms (including abnormal |
| Adverse event | laboratory findings), condition or illness which are not always |
| | related to Humira. |
| | Adverse events which occur from the first administration date of |
| Adverse events in the | Humira through Week 56 of administration (Day 1 + 392) |
| safety analysis period | Note that adverse events in discontinued cases should be the ones |
| salety analysis period | which occur from the first administration date of Humira through |
| | the final administration + 28 days. |
| | Adverse events which occur prior to the first administration date of |
| Adverse events not in the | Humira or beyond Week 56 of administration (Day 1 + 392). |
| safety analysis period | Note that adverse events in discontinued cases should be the ones |
| salety analysis period | which occur prior to the first administration date of Humira or |
| | beyond the final administration + 28 days. |
| Adverse reaction | Adverse events for which the causal relation with Humira cannot be |
| Adverse reaction | ruled out. |
| Adverse reactions in the | Adverse events which occurred in the safety analysis period and for |
| safety analysis period | which the causal relation with Humira cannot be ruled out. |
| Adverse reactions not in | Adverse events which occurred not in the safety analysis period and |
| the safety analysis period | for which the causal relation with Humira cannot be ruled out. |
| | It includes number of cases, mean, standard deviation, minimal |
| Summary statistics | value, 1st quartile value, median, 3rd quartile value and maximal |
| | value. |
| MedDRA/J | Medical Dictionary for Regulatory Activities / Japanese edition |
| SOC | System Organ Class in MedDRA/J |
| PT | Preferred Terms in MedDRA/J |
| LLT | Lowest Level Terms in MedDRA/J |
| IGRA test | Interferon gamma release assay |
| Partial Marya caara | Total of stool frequency sub score, rectal bleeding sub score and |
| Partial Mayo score | physician's global assessment |
| Mayo score | Total of partial Mayo score and endoscopy score |
| GB | Green book. Guide on re-examination |

### 3. Objective of this statistical analysis plan

### 3.1. Objective of developing this statistical analysis plan

This statistical analysis plan aims at planning in advance the items regarding the statistical analysis activities which are conducted in accordance with the protocol of "Special drug-use survey for Humira<sup>®</sup> for subcutaneous use only (the long-term survey on colitis ulcerative)" (hereinafter referred to as "this survey"). This is a survey conducted in accordance with GPSP Ministerial Ordinance, and is a document used to prepare the regulatory report of Humira's special drug-use survey and application documents for re-examination.

### 4. The survey outline

#### 4.1. Survey objective

This survey aims at exploring the following items in colitis ulcerative patients who used Humira, as the special drug-use survey of Humira <sup>®</sup> for subcutaneous use only (the long-term survey).

- 1) Unexpected adverse reactions (Specifically important adverse reactions)
- 2) The onset status of adverse reactions in the practical use
- 3) Factors which may affect the safety and effectiveness

<Priority survey items>

The onset status of infection, tuberculosis, malignant tumour, administration site reactions, autoimmune disease, pancytopenia, demyelinating disease, cardiac failure congestive and interstitial pneumonia

If an intestinal infection occurs, investigate the virus or bacterium causing it whenever possible.

#### 4.2. Survey plan

The patients should have colitis ulcerative in the active moderate or severe phase (only when an existing treatment does not work) and newly receive Humira.

### 4.3. Target sample size for the survey

1500 patients

<Rationale for the sample size>

1. As this survey is conducted in the clinical settings, we expect that the patients with a treatment history with anti-TNFα drugs may be highly observed. Given that the registration of such patients can increase the dropout rate compared to that of the relevant domestic clinical studies, we calculated that the dropout rate would reach 70% at Week 52. Next, given that the number of patients whose CDAI of the effectiveness endpoint was not

provided in the all-case survey for Crohn's disease accounted for approximately 30%, we need 1500 patients with 30% remission rate,  $\pm 5\%$  estimated accuracy of 95% CI and under the conditions where 30% of Mayo score are not assessable (Table 1).

Table 1: The number of patients and accuracy calculated based on the dropout rate

| Dropout rate 70% | | | | |
|------------------|---------|--------------|----------------|-------------|
| | After | Mayo score | At Week 52 | |
| Sample | Week 52 | Number of | Remission rate | A 0011#0017 |
| size | Sample | patients for | 30% | Accuracy |
| | size | assessment | 95%CI | |
| 500 | 150 | 105 | 21.2-38.8 | ±8.8% |
| 1000 | 300 | 210 | 23.8-36.2 | ±6.2% |
| 1500 | 450 | 315 | 24.9-35.1 | ±5.1% |
| 2000 | 600 | 420 | 25.6-34.4 | ±4.4% |

The number of cases with Mayo score provided was calculated as 70% of the total number of patients after Week 52 (i.e., 30% of Mayo score is not provided).

 Next, we examined the accuracy of the remission rate where the number of patients was 1500 as mentioned above with/without treatment experience of anti-TNFα drugs (Table 2).
 We set the following conditions for the accuracy examination:

The all-case survey data in Crohn's-disease patients who used Humira showed that 80% of the patients had been treated with anti-TNF $\alpha$  drugs while 20 % had not. Given that there were many patients who could not benefit from an anti-TNF $\alpha$  agent of prior medication awaiting right after the indication of Crohn's disease was approved, we expect that the same percentage of patients can be enrolled in this survey, too. In this regard, we decided to adopt the similar ratio for the anti-TNF $\alpha$  drug use in this survey and have the patients with and without the treatment history of the drug in an 8:2 ratio.

We set the remission rate of Mayo score at Week 52 in the patients without anti-TNF $\alpha$  drug history as 30% based on the percentage used to estimate the above 1500 patients and in the patients with the history as 10% based on the data in an overseas clinical study (M06-827 Study).

Table 2: The Accuracy of remission rate with/without treatment history of anti-TNFα drugs

| <i>y</i> | | | J | 0 |
|---|---|---|---|---|
| | Mayo score<br>Number of<br>patients for<br>assessment | At Week 52 Remission rate | 95%CI | Accuracy |
| With a treatment history of anti-TNFα drugs | 252 | 10% | 6.1-13.9 | ±3.8% |
| Without a treatment history of anti-TNFα drugs | 63 | 30% | 17.9-42.1 | ±12.1% |

These results suggest that the value might be less accurate due to a fewer number of patients in the group of no treatment history of anti-TNF $\alpha$  drugs while the value in the group with the treatment history will be accurate enough for the examination. (Table 2)

3. For the safety, tuberculosis occurred in a patient (1/177 patients, 0.6%) as an important adverse event (the causal relationship with Humira: probably not related) in a relevant domestic clinical study. If data from 1500 patients are collected based on the incidence, we can assess the accuracy with the 95%CI for the incidence of 0.3%-1.1%. Even if the incidence of tuberculosis reached 2% in this survey, which is higher than that of the clinical study, the confidence interval would range between the minimum 1.35 and the maximum 2.84 by collecting 1500 patients. In this case, the incidence of tuberculosis (as an adverse event) observed in a clinical study for arthritis rheumatoid exceeds 1.0%, meaning that the accuracy is assessable.

Therefore, we have 1500 patients as the target sample size.

### 5. Items to be analyzed and the methods

#### 5.1. Analysis items

- 1) Items regarding patient composition
  - [1] Sample size for registration
  - [2] The number of patients whose survey form was locked
  - [3] The number of patients in the safety analysis group
  - [4] The number of patients in the effectiveness analysis group
- 2) Items regarding safety
  - [1] A list of the onset status of adverse reactions/infections
  - [2] Factors which may affect the safety
    - Incidence of adverse reactions per patient background, etc.
    - Presence/absence of the experience with biological products, and the relation with it
    - Safety for long-term use
    - Safety relationship when anti-adalimumab antibody was measured
    - Presence/absence of self-administration and the relation with it
  - [3] Adverse events which occurred during or after the administration
    - A list of the onset status of serious adverse events, etc.
    - The onset status of intestinal infection of cytomegalovirus colitis
  - [4] Warnings, Careful Administration section, and major adverse events subject to

special attention in Important Precautions section in Humira's package insert (infections including tuberculosis, malignant tumour, injection site reactions, allergic reaction, demyelinating disorders, lupus-like syndrome and blood disorder)

- [5] The administration-error status at self-administration
- [6] The safety in pediatric patients with colitis ulcerative

#### 3) Items regarding effectiveness

- Changes in the effectiveness until Week 52 of administration (Mayo score, partial Mayo score, etc.)
- Presence/absence of the experience with biological products, and the relation with it
- Effectiveness per prior medication history
- Effectiveness for long-term use (including the percentage of the secondary failure)
- Effectiveness relationship when anti-adalimumab antibody was measured
- Effectiveness in pediatric patients with colitis ulcerative

#### 4) Items regarding patients with special backgrounds

A list of onset status of adverse reactions/infections in patients with special backgrounds such as pediatrics, the elderly, pregnant woman, renal impairment, hepatic function disorder, etc.

#### 5.2. Analysis method

Appropriate tests including  $\chi^2$  test are employed for analysis, depending on the analysis-data scale and the characteristics.

### 6. Presence/absence of analysis and its schedule

| Analysis objective | The survey's reporting interval and the deadline |
|---|---|
| | of re-examination |
| The 6th periodical safety | January 1, 2016 to December 31, 2016 |
| report | |
| Re-examination | June 14, 2013 to May 15, 2017 |
| Final report | June 14, 2013 to March 31, 2018 |

# 7. Softwares/dictionary used for analysis

## 7.1. Statistical analysis and listing softwares

The softwares and their versions for use are as follows:

| | Software and version |
|----------------------|-------------------------------------------------------|
| OS | We use Microsoft Windows 7 or a more recent version. |
| Statistical analysis | We use SAS Ver. 9.2 or a more recent version. |
| software | |
| Listing software | We use Microsoft Excel 2010 or a more recent version. |

## 7.2. Dictionary for use

The dictionaries used for the names of adverse events, complications, and drugs are as follows:

| Item | Dictionary and its version | Remarks |
|---|---|---|
| Types of adverse events | Medical Dictionary for Regulatory | They are classified into a |
| and adverse | Activities / Japanese edition | System Organ Class (SOC) and |
| reactions/infections | (MedDRA/J 20.1) | the appropriate term among the |
| | | preferred terms (PT) is selected |
| | | for description. |
| | | SOC is displayed in accordance |
| | | with the international |
| | | agreement. |
| | | The MedDRA/J version used |
| | | will be provided in a blank |
| | | space. |
| Drug name (concomitant | Iyakuhinmei Data File (IDF) *An | • A 7-digit code is used, in |
| medication) | appropriate version should be used | principle, when concomitant |
| | for aggregation, depending on the | medications are counted per |
| | analysis period. | product. |
| | | Give a priority to the lowest |
| | | level codes when using codes |
| | | for the list of concomitant |
| | | medications (including |
| | | Re-examination Attachment |
| | | Form 3). |

# 8. The definition of the groups used for analysis

| Name of group | Definition |
|---|---|
| Registered patients | |
| Patients whose survey | Registered patients whose survey form was locked. |
| form was locked | |
| Patients whose survey | Registered patients whose survey form was yet to be locked. See |
| form was yet to be | Reference Data "Survey form lock/unlock information" for the criteria |
| locked | for the status that a survey form is yet to be locked. |
| Patients excluded from | The patients whose survey form has been locked and who satisfy the |
| the safety analysis group | criteria of the patients excluded from the safety analysis group. See |
| | Reference Data "Inclusion/exclusion of patients" for the criteria to |
| | exclude patients from the safety analysis group. |
| | The exclusion items are as follows: |
| | Breach of contract: unsigned institutions/specialties |
| | Breach of contract: an excess of contracted number of patients |
| | Breach of contract: unsigned physicians |
| | Not treated with Humira |
| | Not confirmed by physician |
| | Overlapped patients |
| | Safety is not assessable |
| | Breach of registration criteria: a deviation from the registration period |
| | Breach of registration criteria: with a history of treatment with |
| | Humira |
| | Administration prior to contract |
| | Data credibility cannot be confirmed: closure/merger of medical |
| | institutions |
| | Data credibility cannot be confirmed: the physician was transferred |
| | Data credibility cannot be confirmed: the physician refuses |
| | confirmation |
| | Data credibility cannot be confirmed: inconsistency was found in the |
| | survey form |
| Patients in the safety | The remaining patients after the patients excluded from the safety |
| analysis group analysis group are removed from the patients whose survey for | |
| | locked |
| Patients excluded from | The patients who satisfy the exclusion criteria for the effectiveness |
| the effectiveness analysis | analysis group. See Reference Data "Inclusion/exclusion of patients" for |

| Name of group | Definition |
|---|---|
| group | the exclusion criteria for the effectiveness analysis group. |
| | The exclusion items are as follows: |
| | Breach of registration criteria: Not the disease to be surveyed |
| | Effectiveness is not assessable |
| Patients in the | The remaining patients after those excluded from the effectiveness |
| effectiveness analysis | analysis group are removed from the patients in the safety analysis |
| group | group. |

# 9. General agreement items for analysis

## 9.1. Handling of missing data

No missing data at any time are imputed for analysis. Note that entry data need to be imputed in some items and the imputation method for imputation-required items is defined in the definitions of each item at Chapter 10 or thereafter.

### 9.2. Descriptive statistics

The following will be calculated for categorial data and quantitative data.

| Data type | Item to be calculated |
|---|---|
| | Number of patients, percentage, etc. |
| | When the percentage is calculated, the number of patients of |
| Catanania 1 data | "unknown" and "not provided" is included in the denominator. Chapter |
| Categorical data | 13 stipulates the details regarding the setting of denominators. |
| | The patients of "unknown" and "not provided" are excluded in the |
| | statistical test. |
| Quantitative data | Number of patients, mean, standard deviation, median, minimal value, |
| | maximal value, etc. |

### 9.3. Display digit for figures

The display digit for figures is as follows:

| Type of figure | Display digit |
|---|---|
| Mean, standard The figure in the significant digit + 2 digits of data is rounded off t | |
| deviation, median | figure in the significant digit of data + 1 digit for display. |
| Minimal value,<br>maximal value | The same number of digits is used for the significant digit of data. |
| Number of patients | Displayed as a whole number |
| | The figure is rounded off to the nearest one decimal place for display. |
| Percentage, 95% | When figures for Attachment Form 2, incidences of adverse events, etc are |
| Confidence Interval | rounded off to two decimal places, the details are specified in the chart |
| | layout. |
| | Round the 5 decimal places down to the 4 decimal places. |
| p value | When the figure is smaller than 0.0001, display it as <0.0001 across the |
| | board. |
| | The figure for duration of illness should be displayed with the significant |
| | digit rounded to the one decimal place. |
| Significant digit | For others, the display digit of data should be the significant digit. |
| | As for CRP, the summary statistics except the number of patients should |
| | be rounded off to two decimal places. |

### 9.4. Figure display rule

| Case | Display rules |
|----------------|---------------|
| If a figure is | Hyphen "-" |
| incalculable | |

#### 9.5. Statistical test method

The test does not include the classification of unknown/not provided. In principle, the first layer is subjected to the intersegmental test of classified data. When adjusting multiplicity, describe it in each chart of Chapter 13.

### 9.6. Significant level

In principle, the significant level is 5%, two-tailed. p<0.05 (<5%) shall be considered significant.

# 10. Derivation and calculation methods for data

## 10.1. General

| Data name | Derivation and calculation methods |
|---|---|
| | If the same code is found among the DCF codes of "[Humira |
| Number of site | UC]DCF code list_Company A" "[Humira UC]DCF code |
| | list_Company E", it should be regarded as 1 site. |
| Number of patients per | The number of patients are calculated per the identical DCF site |
| site | code. |
| Patients with an adverse | |
| event which occurred not | Patients with at least one adverse event which occurred not in the |
| in the safety analysis | safety analysis period |
| period | |
| Patients who developed | Patients with at least one event which is categorized into infection in |
| an infection | the "Priority Survey Item List_MedDRA20.1_FIX". |
| Patients who developed | Patients with at least one event which is categorized into tuberculosis |
| tuberculosis | in the "Priority Survey Item List_MedDRA20.1_FIX". |
| Patients who developed | Patients with at least one event which is categorized into malignant |
| malignant tumour | tumour in the "Priority Survey Item List_MedDRA20.1_FIX". |
| Patients who developed | Patients with at least one event which is categorized into |
| an administration site | administration site reaction in the "Priority Survey Item |
| reaction | List_MedDRA20.1_FIX". |
| Patients who developed | Patients with at least one event which is categorized into |
| an autoimmune disease | auto-immune disease in the "Priority Survey Item |
| an autominune disease | List_MedDRA20.1_FIX". |
| Patients who developed | Patients with at least one event which is categorized into |
| pancytopenia | pancytopenia in the "Priority Survey Item List_MedDRA20.1_FIX". |
| Patients who developed | Patients with at least one event which is categorized into |
| demyelinating disease | demyelinating disease in the "Priority Survey Item |
| demyelmating disease | List_MedDRA20.1_FIX". |
| Patients who developed | Patients with at least one event which is categorized into cardiac |
| cardiac failure | failure congestive in the "Priority Survey Item |
| congestive | List_MedDRA20.1_FIX". |
| Patients who developed | Patients with at least one event which is categorized into interstitial |
| interstitial pneumonia | pneumonia in the "Priority Survey Item List_MedDRA20.1_FIX". |
| Patients subject to AAA | Patients who are described in "UC Survey AAA Measurement (final |
| measurement | report)". |

| Data name | Derivation and calculation methods |
|---|---|
| | administration date. If the next record has already been generated and the first administration date of the next record comes earlier than the date imputed as the final date |
| | of the year, impute the first administration date of the next record - 1 day for the final administration date. |
| | Of note, if the final administration date is provided in the record where the final administration date of Humira has been identified according to the above rule and the "continued" checkbox is checked, follow the below: |
| | <ul> <li>If the described final administration date &gt; the final administration date imputed according to the above rule, select the imputed final administration date as the final administration date of Humira for the patient.</li> <li>If the described final administration date &lt;= the final administration date imputed according to the above rule, select the described final administration date as the final administration date of Humira for the patient.</li> </ul> |
| | If the first administration date of Humira + 364 days < the final administration date of Humira imputed according to the above rule, select the first administration date of Humira + 364 days as the final administration date of Humira. |
| Days to the final administration date of Humira | The final administration date of Humira - the first administration date of Humira + 1 |
| Administration status (dosage and administration) | Sort the data by the first administration date provided in "the administration status of Humira" in the survey form and aggregate the administration status (dosage and administration) according to the following rules: • If all the following [1] to [4] are satisfied, aggregate the data as "160mg→80mg→40mg once every two weeks and no changes thereafter". • If none of the following [1] to [4] is satisfied Aggregate as "others". [1] 1st administration: as a patient with a dose of 160mg |

| Data name | Derivation and calculation methods |
|---|---|
| | [2] 2nd administration: as a patient with a dose of 80mg |
| | [3] 3rd administration and thereafter: the dosing |
| | frequency "once every 2 weeks" is checked in the |
| | survey form, and a patient with a dose of 40mg |
| | * If the patient receives the third administration and |
| | thereafter, all the administration status should be the |
| | condition as shown in [3]. |
| | [4] Patients who did not have a washout period for 30 |
| | days or longer. |
| | If the administration status (dose and administration) is categorized |
| | in "others", follow the rules below to find the reason for the change |
| | in dose/dosing frequency. |
| | • 1st dose: "a reason for other than 160mg (a dose) or in the |
| | case of self-administration" in the survey form. |
| Reason for change in | • 2nd dose: "a reason for other than 80mg (a dose) or in the case |
| dose/dosing frequency | of self-administration" in the survey form. |
| | • 3rd and the subsequent dose(s): "a reason for other than 40mg |
| | (a dose), or in the case of other than once every 2 weeks |
| | (dosing frequency)" or "reason for change in dose/dosing |
| | frequency" in the survey form. |
| | Dosing frequency |
| | [1] Sort data in the order of "the first administration date" of "the |
| | administration status of Humira", dosing frequency and |
| | description. |
| | [2] Calculate the dosing interval per data on administration status |
| | The interval between first and second administrations should |
| Administration status | be 14 days. |
| | • For the third and subsequent dose(s), the interval should be 14 |
| (total number of dosing, | days if the dosing frequency "once every 2 weeks" is checked |
| total dose) | while the dosing frequency should be obtained from "[Humira |
| | UC] Conversion data provided for analysis" if the dosing |
| | frequency is "others". |
| | [3] Calculate the dosing frequency per data on administration |
| | status. |
| | Dosing frequency = (the final administration date (after |
| | imputed) – the first administration date(after imputed))/dosing |

| Data name | Derivation and calculation methods |
|---|---|
| | frequency (number of days) |
| | [4] When the results of [3] are ">0" (bigger than 0) and "<1" |
| | (smaller than 1), the dosing frequency shall be counted as 1. |
| | If the figure is ">=1" (1 or bigger), round the decimal down to the |
| | integer for the dosing frequency. |
| | [5] The total number of dosing shall be the total of [4] per patient. |
| | • Dose |
| | [1] If "Others" of a Humira dose is checked, the dose should be |
| | obtained from "[Humira UC] Conversion data provided for |
| | analysis". |
| | [2] Calculate the dose per data of the administration status. |
| | Dose = the number of dosing * a dose |
| | [3] The total dose should be the total of [2] per patient. |
| | • The mean daily dose |
| | The mean daily dose = the total dose/the total number of dosing |
| | If a patient's final administration date of Humira comes before the |
| | first administration date of Humira + 336, we handle the patient as a |
| Discontinued patients | discontinued case. |
| | Follow the above definition, no matter whether the discontinuation is |
| | selected in the survey form. |
| | "Present" is defined for the situation where a patient qualifies for the |
| | defined discontinued case and at least one has been checked in |
| Presence/absence of | "reason for discontinuation" of "discontinuation of the survey" of the |
| reason for | survey form. On the other hand, if a patient qualifies for the defined |
| discontinuation | discontinued case and no description has been made in the "reason |
| | for discontinuation" column in the survey form, the case is defined as |
| | an "unknown/not provided" case. |
| | It should derive from "reason for discontinuation" of |
| Reason for | "discontinuation of the survey" of the survey form. Recode the |
| discontinuation | reason for discontinuation based on other descriptions of "reason for |
| discontinuation | discontinuation" and "[Humira UC] Conversion data provided for |
| | analysis". Select "unknown/not provided" for undescribed data". |
| Reason for | Obtain the detailed items of reason for discontinuation "others" in |
| discontinuation, other | "[Humira UC] Conversion data provided for analysis". |
| reasons | |
| Patients who continue | The patients who are not the discontinued cases are regarded as the |

| Data name | Derivation and calculation methods |
|---|---|
| the survey | patients who continue the survey |
| Presence/absence of | When complication data are contained in the survey form, it should |
| | be classified as "with complications". When there is no description of |
| | "presence/absence of complications" in the survey form or the |
| complications | assessment is impossible, it should be classified as "unknown/not |
| | provided", and other cases are "no complications". |
| | When medical-history data are contained in the survey form, it |
| Presence/absence of | should be classified as "with medical history". When there is no |
| | description of "presence/absence of medical history" in the survey |
| medical history | form or the assessment is impossible, it should be classified as |
| | "unknown/not provided", and other cases are "no medical history". |
| Complication/Hepatic | When hepatic function disorder data are contained in "171210 |
| function disorder | Complication", it should be classified as "with hepatic function |
| Tunction disorder | disorder". other cases are "no hepatic function disorder". |
| Complication/Renal | When renal impairment data are contained in "171210 |
| impairment | Complication", it should be classified as "with renal impairment". |
| шрантен | other cases are "no renal impairment". |
| Presence/absence of | When circulatory disorder data are contained in "171210 |
| Complication/Circulator | Complication", it should be classified as "with circulatory disorder". |
| y disorder | other cases are "no circulatory disorder". |
| Presence/absence of | When blood disorder data are contained in "171210 Complication", it |
| Complication/Blood | should be classified as "with blood disorder. Other cases are "no |
| disorder | disorder". |
| Presence/absence of | When respiratory disorder data are contained in "171210 |
| Complication/Respiratory | Complication", it should be classified as "with respiratory disorder. |
| disorder | Other cases are "no respiratory disorder". |
| | If a survey form contains the data other than hepatic function |
| | disorder, renal impairment, circulatory disorder, blood disorder and |
| | respiratory disorder, it should be classified as "with other |
| | complications". Others are "no other complications". |
| Presence/absence of | |
| Complication/others | If a survey form contains the data in "171210 Complication" for |
| | presence/absence of diabetes mellitus, gastrointestinal disorder, |
| | osteoporosis and malignant tumour as well among the detailed |
| | classifications of other complications, it should be classified as "with |
| | complications". Others are "no complications". |

| Data name | Derivation and calculation methods |
|---|---|
| | If a survey form contains the data on complications other than |
| | diabetes mellitus, gastrointestinal disorder, osteoporosis and |
| | malignant tumour among the detailed classifications of other |
| | complications, it should be classified as "with other complication of |
| | other detailed classifications". Others are "no other complication of |
| | other detailed classifications". |
| | As for collagen disorder, if "other: collagen disorder" in |
| | "complications" of "patient information" is checked, it should be |
| | classified as "with collage disorder. Other cases are "no collagen |
| | disorder". |
| Medical history: | When tuberculosis data are contained in "180111 Medical history", it |
| presence/absence of | should be classified as "with tuberculosis. Other cases are "no |
| tuberculosis | tuberculosis". |
| Medical history: | When non-tuberculous mycobacteriosis data are contained in |
| presence/absence of | "180111 Medical history", it should be classified as "with |
| non-tuberculous | non-tuberculous mycobacteriosis. Other cases are "no |
| mycobacteriosis | non-tuberculous mycobacteriosis". |
| Medical history: | When interstitial pneumonia data are contained in "180111 Medical |
| presence/absence of | history", it should be classified as "with interstitial pneumonia. Other |
| interstitial pneumonia | cases are "no interstitial pneumonia". |
| Medical history: | When bronchitis bacterial data are contained in "180111 Medical |
| presence/absence of | history", it should be classified as "with bronchitis bacterial. Other |
| bronchitis bacterial | cases are "no bronchitis bacterial". |
| Medical history: | When aplastic anaemia data are contained in "180111 Medical |
| presence/absence of | history", it should be classified as "with aplastic anaemia. Other |
| aplastic anaemia | cases are "no aplastic anaemia". |
| Medical history: | When pancytopenia data are contained in "180111 Medical history", |
| presence/absence of | it should be classified as "with pancytopenia. Other cases are "no |
| pancytopenia | pancytopenia". |
| Medical history: | When malignant tumour data are contained in "180111 Medical |
| presence/absence of | history", it should be classified as "with malignant tumour. Other |
| malignant tumour | cases are "no malignant tumour". |
| Medical history: | When medical-history data except tuberculosis, non-tuberculous |
| presence/absence of | mycobacteriosis, interstitial pneumonia, bronchitis bacterial, aplastic |
| other medical history | anaemia, pancytopenia and malignant tumour are contained among |
| other medical history | the medical-history data in the survey form, it should be classified as |

| Data name | Derivation and calculation methods |
|---|---|
| | "with other medical history". The remaining cases are "no other |
| | medical history". |
| | When "with allergy history in "patient information" of the survey |
| | form is checked, it should be classified as "with allergy history. |
| Presence/absence of | When "allergy history unknown" is checked, it should be "unknown" |
| allergy history | whereas nothing is provided in "presence/absence of allergy history" |
| | of the form, it should be "not provided". Other cases are "no allergy |
| | history". |
| | When "Hepatitis→viral" is selected in "Complications" of "Patient |
| | information" in the survey form and also "B" is selected for |
| Patients with an hepatitis | "Hepatitis virus carrier", the patient is classified as a patient with an |
| B virus infection | hepatitis B virus infection. The patients also include those developed |
| | an adverse event encoded with the applicable MedDRA PT described |
| | in "patients with 180111B Hepatitis B virus infection". |
| | For the items for smoking history in the survey form, when the |
| | checkboxes of "smoking" or "in the past" are checked, or when "with |
| | smoking history" is checked and the smoking period is "unknown", |
| Presence/absence of | both cases should be classified as "with smoking history". When |
| smoking history | "unknown" is checked for smoking history, it should be "unknown". |
| | When nothing is described in "presence/absence of smoking history" |
| | of the survey form, it should be "not provided". |
| | Other cases are "no smoking history". |
| | When "smoking" is checked among the items for smoking history in |
| | the survey form, or when any descriptions are made in the smoking |
| | period of "smoking", they should be classified as "smoking". When |
| Detailed classification of | "in the past" is checked or any descriptions are made in the smoking |
| | period "in the past" in patients who are not classified as "smoking", |
| smoking history | the case should be classified as "only in the past (not smoking now)". |
| | When "with smoking" is checked but nothing is checked in the |
| | detailed classification, or when "unknown" is checked, they should |
| | be "unknown". |
| Patients with dosing | Patients other than those who satisfied [1] to [4] of "Administration |
| deviation of Humira | status (dosage and administration)" |
| Presence/absence of | When "Self-administration" in the "Administration status of Humira" |
| self-administration | column is checked at least once, the case should be classified as |
| | "with" self-administration. Others are "without" self-administration. |

| Data name | Derivation and calculation methods |
|---|---|
| | When both "administration by physician" and "self-administration" |
| | are checked, the case should be "with self-administration". |
| | When "with" self-administration error is checked in the survey form, |
| | it should be classified as "with" the error. When "without" is |
| D / 1 C | checked, it should be "without" the error. |
| Presence/absence of | When some details are provided along with the onset date in the |
| self-administration error | self-administration error column irrespective of a check on |
| | "with"/"without", it should be regarded as "with" the error. |
| | If nothing is described there, it should be "unknown/not provided". |
| | It should be identified based on the sex in the patient's information of |
| G. | the survey form. When multiple items are checked or data without a |
| Sex | description are included, the case should be classified as |
| | "unknown/not provided". |
| | It should be identified based on pregnancy/nursing in the patient's |
| | information of the survey form. When multiple items are checked or |
| <b>.</b> | data without a description are included even if the sex has been |
| Pregnancy/nursing | selected as "woman", the case should be classified as "unknown/not |
| | provided". If the sex is not "woman" even though a description has |
| | been made for this item, it is excluded from the calculation. |
| | It should be identified based on the race in the registration form. |
| Race | When multiple items are checked or data without a description are |
| | included, the case should be classified as "unknown/not provided". |
| | It should be identified based on the year and month of the patient's |
| | birth or the first administration date of Humira in the survey form. |
| | For the date of birth, the first day should be imputed to identify it, |
| | using the following SAS code. |
| | floor((intck('month', date of birth, the first administration date of |
| A | Humira) - (day(the first administration date of Humira) < day(date of |
| Age | birth)))/12) |
| | Of note, if it is impossible to identify the date of birth or the first |
| | administration date of Humira due to an incomplete or unknown date, |
| | select the age provided in the survey form. |
| | If it cannot be identified based on the date of birth or the age is not |
| | provided, it is defined as "unknown/not provided". |
| Pediatrics | Patients aged <15 years |
| The elderly | Patients aged ≥65 years |

| Data name | Derivation and calculation methods |
|---|---|
| Body weight | It should be identified based on the body weight in the patient's |
| | information of the survey form. When "unknown" is checked or data |
| | without a description are included, it should be "unknown/not |
| | provided". |
| | It should be identified based on the height in the patient's information |
| Body height | of the survey form. When "unknown" is checked or data without a |
| | description are included, it should be "unknown/not provided". |
| BMI | Body weight (kg) / (Body height (cm)/100) <sup>2</sup> |
| | "For XX years and XX months" should be converted into the figure |
| | in years for "duration of illness" of "patient information" in the |
| | survey form. |
| Duration of illness (in | When both figures of year and month: year + month/12 |
| years) | When the figure of year is provided: year |
| | When the figure of month is provided: month/12 |
| | Other cases are identified as "unknown/not provided" as the duration |
| | cannot be identified. |
| | If both "colitis ulcerative" and "others" are checked for indication in |
| Indication | the survey form, it should be calculated as "colitis ulcerative". |
| | It should be identified based on "site of disease of colitis ulcerative" |
| Site of disease | in the survey form. Select "unknown/not provided" for undescribed |
| | data". |
| | Conducted: When "HBs antigen test" in the survey form was |
| | conducted (If "conducted" was not checked but the test results were |
| IIDa antigan taat | provided, it should be regarded as "conducted") |
| HBs antigen test | Not conducted: When "HBs antigen test" in the survey form was not |
| | conducted |
| | Unknown/not provided: other than the above |
| | Conducted: When "HBs antibody test" in the survey form was |
| | conducted (If "conducted" was not checked but the test results were |
| HBs antibody test | provided, it should be regarded as "conducted") |
| | Not conducted: When "HBs antibody test" in the survey form was |
| | not conducted |
| | Unknown/not provided: other than the above |
| | Conducted: When "HBc antibody test" in the survey form was |
| HBc antibody test | conducted (If "conducted" was not checked but the test results were |
| | provided, it should be regarded as "conducted") |

| Data name | Derivation and calculation methods |
|---|---|
| | Not conducted: When "HBc antibody test" in the survey form was |
| | not conducted |
| | Unknown/not provided: other than the above |
| | Conducted: When "HBV-DNA quantification assay" in the survey |
| | form was conducted (If "conducted" was not checked but the assay |
| HBV-DNA | results were provided, it should be regarded as "conducted") |
| quantification assay | Not conducted: Not conducted: When "HBV-DNA quantification |
| | assay" in the survey form was not conducted |
| | Unknown/not provided: other than the above |
| | Conducted: When either of "Tuberculin test" or "IGRA" was |
| | conducted (If "conducted" was not checked but the results were |
| Tuberculin test or IGRA | provided, it should be regarded as "conducted") |
| Tuberculin test of IGRA | Not conducted: When neither "Tuberculin test" nor "IGRA" was |
| | conducted |
| | Unknown/not provided: other than the above |
| | When the first administration date of Humira is 1 and a day before |
| | the first administration date is -1, the patients who underwent chest X |
| Chest X ray test | ray test should have a record in which the chest X ray test was |
| | conducted between -90 and 1. Of note, the data in the survey form |
| | shall be used. |
| | When the first administration date of Humira is 1 and a day before |
| | the first administration date is -1, the patients who underwent |
| Chest CT test | thoracic CT test should have a record in which the CT test was |
| | conducted between -90 and 1. Of note, the data in the survey form |
| | shall be used. |
| | When the first administration date of Humira is 1 and a day before |
| | the first administration date is -1, the patients who underwent any |
| Other imaging | other imaging should have a record in which the imaging was |
| | conducted between -90 and 1. Of note, the data in the survey form |
| | shall be used. |
| | Conducted: When either "chest X ray" or "CT test" in the survey |
| Chest X ray or CT test | form was conducted (If "conducted" was not checked but the test |
| | results were provided, it should be regarded as "conducted") |
| | Not conducted: other than the above |
| Presence/absence of prior | The drug names described in "prior-medication history for colitis |
| medications | ulcerative" in the survey form should be regarded as the prior |

| Data name | Derivation and calculation methods |
|---|---|
| | medications. Note that when a drug code is null, it is not regarded as a prior medication. When prior-medication data are contained in the survey form, it |
| Presence/absence of prior medication (aminosalicylic acid | when prior-medication data are contained in the survey form, it should be classified as "with prior medication". When there is no description of "presence/absence of prior medications" in the survey form or the assessment is impossible, it should be classified as "unknown/not provided", and other cases are "without prior medications". Refer to "171218 drug list_UC". If prior-medication data of the applicable drug code are provided in the survey form, or if an aminosalicylic acid drug in the survey form is checked, regard the case as "with aminosalicylic acid". Others are "without |
| drug) | aminosalicylic acid". Refer to "171218 drug list UC". If prior-medication data of the |
| Presence/absence of prior medication (corticosteroids) | applicable drug code are provided in the survey form, or if corticosteroids in the survey form is checked, regard the case as "with corticosteroids". Others are "without corticosteroids". |
| Presence/absence of prior medication (azathioprine) | Refer to "171218 drug list_UC". If prior-medication data of the applicable drug code are provided in the survey form, or if azathioprine in the survey form is checked, regard the case as "with azathioprine". Others are "without azathioprine". |
| Presence/absence of prior medication (6-mercaptopurine) | Refer to "171218 drug list_UC". If prior-medication data of the applicable drug code are provided in the survey form, or if 6-mercaptopurine in the survey form is checked, regard the case as "with 6-mercaptopurine". Others are "without 6-mercaptopurine". |
| Presence/absence of prior medication (azathioprin & 6-mercaptopurine) | Refer to "171218 drug list_UC". If prior-medication data of the applicable drug code are provided in the survey form, or if azathioprin and 6-mercaptopurine in the survey form are checked, regard the case as "with azathioprin & 6-mercaptopurine". Others are "without azathioprin & 6-mercaptopurine". |
| Presence/absence of prior medication (tacrolimus & ciclosporin) | Refer to "171218 drug list_UC". If prior-medication data of the applicable drug code are provided in the survey form, or if tacrolimus & ciclosporin in the survey form is checked, regard the case as "with tacrolimus & ciclosporin". Others are "without tacrolimus & ciclosporin". |
| Presence/absence of | Refer to "171218 drug list_UC". If prior-medication data of the |
| Data name | Derivation and calculation methods |
|---|---|
| prior medication | applicable drug code are provided in the survey form, or if antibiotics |
| (antibiotics) | in the survey form is checked, regard the case as "with antibiotics". |
| | Others are "without antibiotics". |
| | When any items other than biological products in the survey form are |
| | checked, and when prior medication data on the drug code applicable |
| Presence/absence of | to the drug other than aminosalicylic acid drug, corticosteroids, |
| prior medication (others) | azathioprine, 6-mercaptopurine, tacrolimus, ciclosporin and |
| | antibiotics are included in reference to "171218 drug list_UC", |
| | regard it as "with others". Other cases are "without others". |
| Presence/absence of | Refer to "171218 drug list_UC". If prior-medication data of the |
| | applicable drug code are provided in the survey form, or if Infliximab |
| prior medication (Infliximab) | in the survey form is checked, regard the case as "with Infliximab". |
| (IIIIIXIIIIau) | Others are "without Infliximab". |
| | When 'biological products' is checked in the survey form, and when |
| Presence/absence of | prior-medication data of the drug codes other than Infliximab are |
| prior medication (other | provided in the survey form in reference to "171218 drug list_UC", |
| biological products) | regard the case as "with other biological products". Others are |
| | "without other biological products". |
| | The cases with either "with prior medication (Infliximab)" or "with |
| | prior medication (other biological products)" are regarded as "with a |
| Presence/absence of | treatment history with biological products". Others are "without a |
| treatment history with | treatment history with biological products". |
| biological products | As for presence/absence of the history by 'detailed classification |
| biological products | "with" biological products', if the applicable data among |
| | "Infliximab" and "other biological products" are contained, the case |
| | is regarded as "with" the history. Others are "without" the history. |
| | When the description is made in "Prior treatment for colitis ulcerative |
| | (including surgery)" of the survey form, regard it as a prior treatment. |
| Dungan og/ohannon of | When prior-treatment data are contained in the survey form, it should |
| Presence/absence of prior treatment | be classified as "with prior treatment". When there is no description |
| | of "presence/absence of prior treatment" in the survey form or the |
| | assessment is impossible, it should be classified as "unknown/not |
| | provided", and other cases are "without prior treatment". |
| Draganaa/ahaanaa af | Surgery should be selected if the checkbox of prior treatment |
| Presence/absence of | (surgery) in "prior treatment for colitis ulcerative (including |
| prior treatment (surgery) | surgery)" is checked and if any prior treatment considered as surgery |

| Data name | Derivation and calculation methods |
|---|---|
| | is included in "[Humira UC] Conversion data provided for analysis". |
| | When the data applicable to surgery are contained, regard it as "with |
| | surgery". Others are "without surgery". |
| | If "leukocytapheresis" in "prior treatment (including surgery) for |
| Presence/absence of | colitis ulcerative" is checked and it is not applicable to with prior |
| prior treatment | treatment (surgery) in the survey form, it shall be classified into |
| (leukocytapheresis) | "with leukocytapheresis". Other cases are "without |
| | leukocytapheresis". |
| | If "enteral nutrition therapy" in "prior treatment (including surgery) |
| Presence/absence of | for colitis ulcerative" is checked and it is not applicable to with prior |
| prior treatment (enteral | treatment (surgery) in the survey form, it shall be classified into |
| nutrition therapy) | "with enteral nutrition therapy". Other cases are "without enteral |
| | nutrition therapy". |
| Presence/absence of | If "intravenous nutrition therapy" in "prior treatment (including |
| | surgery) for colitis ulcerative" is checked and it is not applicable to |
| prior treatment | with prior treatment (surgery) in the survey form, it shall be classified |
| (intravenous nutrition | into "with intravenous nutrition therapy". Other cases are "without |
| therapy) | intravenous nutrition therapy". |
| Presence/absence of | If "other therapy" in "prior treatment (including surgery) for colitis |
| | ulcerative" is checked and it is not applicable to with prior treatment |
| prior treatment (other | (surgery) in the survey form, it shall be classified into "with other |
| therapy) | therapy". Other cases are "without other therapy". |
| | Concomitant medications should the data satisfying the following |
| | rules: Note that when a drug code is null, it is not regarded as a |
| | concomitant medication. |
| | When concomitant-medication data are contained in the survey form, |
| | it should be classified as "with concomitant medications". When |
| | there is no description of "presence/absence of prior/concomitant |
| Presence/absence of | medications" in the survey form or the assessment is impossible, it |
| concomitant medication | should be classified as "unknown/not provided", and other cases are |
| | "without concomitant medications". |
| | ◆ Data with drug names in "the administration status of |
| | prior/concomitant medications for colitis ulcerative", "the |
| | administration status of other concomitant medication" of the survey |
| | form. |

| Data name | Derivation and calculation methods |
|---|---|
| Data name | <ul> <li>Derivation and calculation methods</li> <li>When the year and month are described for the first administration date of the concomitant medication, impute "1" for the "date".</li> <li>When the year is described for the first administration date of the concomitant medication, impute "1" each for the "month" and "date".</li> <li>When the year and month are described for the final administration date of the concomitant medication, impute the month's final date for the date.</li> <li>When the year is described for the final administration date of the concomitant medication, impute "12" for the month and "31" for the date.</li> <li>When the final administration of concomitant medication &lt; the first administration date of Humira, and/or when the final administration date of Humira &lt; the first administration date of concomitant medication. If the above imputing methods do not help add the date (the first administration date or the final administration date is not provided, etc.), or if the first administration date of concomitant medication are reversed, it should be regarded as a</li> </ul> |
| | <ul> <li>Data with drug names in "priortreatment history for colitis ulcerative" of the survey form</li> <li>When the year and month are described for the first administration date of the prior medication, impute "1" for the "date".</li> <li>When the year is described for the final administration date of the prior medication, impute "1" each for the month and the date.</li> <li>If the final administration date of the prior medication ≥ the first administration date of Humira, regard it as a concomitant medication. If the above imputing methods do not help add the date, the final administration date of the prior medication shall be unknown and the case should not be regarded as a concomitant medication.</li> </ul> |

| Data name | Derivation and calculation methods |
|---|---|
| | ◆ Data with a drug name in "administration status of |
| | anti-tuberculosis drug" of the survey form |
| | When the year and month are described for the first |
| | administration date of anti-tuberculosis drug, impute "1" for the "date". |
| | When the year is described for the first administration date of |
| | anti-tuberculosis drug, impute "1" each for the "month" and "date". |
| | When the year and month are described for the final |
| | administration date of anti-tuberculosis drug, impute the |
| | month's final date for the date. |
| | When the year is described for the final administration date of |
| | anti-tuberculosis drug, impute "12" for the month and "31" for the date. |
| | When the final administration of anti-tuberculosis drug < the |
| | first administration date of Humira, and/or when the final |
| | administration date of Humira < the first administration date of |
| | anti-tuberculosis drug, exclude the case from the calculation for |
| | concomitant medication. If the above imputing methods do not |
| | help add the date (the first administration date or the final |
| | administration date is not provided, etc.), or if the first |
| | administration date and the final administration date of |
| | anti-tuberculosis drug are reversed, it should be regarded as a concomitant medication. |
| | concomitant medication. |
| | ('Clear' refers to a condition where no ambiguous expressions |
| | like "around", "in the middle", etc. are included and a number |
| | of figure only is provided.) |
| Presence/absence of | Refer to "171218 drug list_UC". If concomitant-medication data of |
| concomitant medication | the applicable drug code are provided in the survey form, regard the |
| (aminosalicylic acid | case as "with aminosalicylic acid". Others are "without |
| drug) | aminosalicylic acid". |
| Presence/absence of | Refer to "171218 drug list_UC". If concomitant-medication data of |
| concomitant medication | the applicable drug code are provided in the survey form, regard the |
| (corticosteroids) | case as "with corticosteroids". Others are "without corticosteroids". |
| Presence/absence of | Refer to "171218 drug list_UC". If concomitant-medication data of |

| Data name | Derivation and calculation methods |
|---|---|
| concomitant medication | the applicable drug code are provided in the survey form, regard the |
| (azathioprine) | case as "with azathioprine". Others are "without azathioprine". |
| Presence/absence of concomitant medication (6-mercaptopurine) Presence/absence of concomitant medication | Refer to "171218 drug list_UC". If concomitant-medication data of the applicable drug code are provided in the survey form, regard the case as "with 6-mercaptopurine". Others are "without 6-mercaptopurine". Refer to "171218 drug list_UC". If concomitant-medication data of the applicable drug code are provided in the survey form, regard the |
| (azathioprine & | case as "with azathioprine & 6-mercaptopurine". Others are "without |
| 6-mercaptopurine) Presence/absence of concomitant medication (tacrolimus & ciclosporin) | azathioprine & 6-mercaptopurine". Refer to "171218 drug list_UC". If concomitant-medication data of the applicable drug code are provided in the survey form, regard the case as "with tacrolimus & ciclosporin". Others are "without tacrolimus & ciclosporin". |
| Presence/absence of | Refer to "171218 drug list UC". If concomitant-medication data of |
| concomitant medication (antibiotics) | the applicable drug code are provided in the survey form, regard the case as "with antibiotics". Others are "without antibiotics". |
| Presence/absence of concomitant medication (others) | When concomitant-medication data on the drug code applicable to the drug other than aminosalicylic acid drug, corticosteroids, azathioprine, 6-mercaptopurine, tacrolimus, ciclosporin and antibiotics are included in reference to "171218 drug list_UC", regard it as "with others". Other cases are "without others". |
| Presence/absence of<br>administration of<br>anti-hepatitis B virus<br>agent | If the following drug codes are included in the survey form, regard the case as "with administration of an anti-hepatitis B virus agent". Others are "without administration of an anti-hepatitis B virus agent". Entecavir (Baraclude): 6250029 Tenofovir (Tenozet, Viread): 6250024 Adefovir (Hepsera): 6250026 Lamivudine: 6250006, 6250020 |
| Presence/absence of concomitant therapy | It should be described in "non-medicinal treatment/concomitant therapy (including surgery) for colitis ulcerative" of the survey form. The data from the first administration date to the final administration date of Humira will be calculated. Such data are also subject to calculation even if the first/final administration dates of concomitant treatment are not unknown. (Only when the days are not overlapped with the administration |

| Data name | Derivation and calculation methods |
|---|---|
| | period of Humira, they shall be excluded from the calculation.) When |
| | concomitant-therapy data are contained in the survey form, it should |
| | be classified as "with concomitant therapy". When "presence/absence |
| | of prior/concomitant medications" is not provided in the survey form |
| | or the assessment is impossible, it should be classified as |
| | "unknown/not provided", and other cases are "without concomitant |
| | therapy". |
| | Surgery should be selected when the 'surgery' checkbox of |
| | non-medicinal treatment/concomitant therapy name is checked in |
| D /1 C | "non-medicinal treatment/concomitant therapy for colitis ulcerative |
| Presence/absence of | (including surgery)" and when any concomitant therapy considered |
| concomitant therapy | as surgery is included in "[Humira UC] Conversion data provided for |
| (surgery) | analysis". |
| | When the data applicable to surgery are contained, regard it as "with |
| | surgery". Others are "without surgery". |
| | If "leukocytapheresis" in "non-medicinal treatment/concomitant |
| Presence/absence of | therapy (including surgery) for colitis ulcerative" is checked and it is |
| concomitant therapy | not applicable to with concomitant therapy (surgery) in the survey |
| (leukocytapheresis) | form, it shall be classified into "with leukocytapheresis". Other cases |
| | are "no leukocytapheresis". |
| | If "enteral nutrition therapy" in "non-medicinal |
| Presence/absence of | treatment/concomitant therapy (including surgery) for colitis |
| concomitant therapy | ulcerative" is checked and it is not applicable to with concomitant |
| (enteral nutrition | therapy (surgery) in the survey form, it shall be classified into "with |
| therapy) | enteral nutrition therapy". Other cases are "no enteral nutrition |
| | therapy". |
| | If "intravenous nutrition therapy" in "non-medicinal |
| Presence/absence of | treatment/concomitant therapy (including surgery) for colitis |
| concomitant therapy | ulcerative" is checked and it is not applicable to with concomitant |
| (intravenous nutrition | therapy (surgery) in the survey form, it shall be classified into "with |
| therapy) | intravenous nutrition therapy". Other cases are "no intravenous |
| | nutrition therapy". |
| Presence/absence of | If "other therapy" in "non-medicinal treatment/concomitant therapy |
| concomitant therapy | (including surgery) for colitis ulcerative" is checked and it is not |
| (other therapy) | applicable to with concomitant therapy (surgery) in the survey form, |
| (other therapy) | it shall be classified into "with other therapy". Other cases are "no |

| Data name | Derivation and calculation methods |
|---|---|
| | other therapy". |
| Tuberculosis test | Conducted: when both "Tuberculin test or IGRA" and "Chest X ray |
| | or CT test" were conducted |
| | Not conducted: other than the above |
| | Conducted: when "HBV-DNA quantification assay" in the survey |
| Hepatitis B test | form was conducted, or |
| | when the results are negative in HBs antigen test, HBs antibody test, |
| | and HBc antibody test. |
| | Not conducted: other than the above |

## 10.2. Safety analysis

| Data name | Derivation and calculation methods |
|---|---|
| | The adverse events for analysis should include not only the events derived |
| | from the survey form but also the events covered in the detailed |
| | investigation which has been described by the physicians at a contracted |
| | site/department even though not derived from the survey form in "AE |
| | matching results". |
| Adverse event | With adverse event: at least 1 record on adverse event(s) exists |
| | Without adverse event: other than the above. |
| | When adverse events are counted per SOC, the identical SOC in a patient |
| | should be counted as 1 whereas the same PT in the same patient be |
| | counted as 1 for PT. When no applicable patients were observed, display |
| | "0" for the number of patients and "0.00" for the percentage. |
| | Based on the seriousness criteria for company assessment which are |
| | provided in "AE matching results", regard the events which have been |
| | assessed to be serious as serious adverse events. |
| Seriousness of | With serious adverse event: at least 1 record on serious adverse event(s) |
| adverse events | exists |
| | Without serious adverse event: other than the above. |
| | Follow the way of counting adverse events to count serious adverse |
| | events. |
| | All events which are not determined as "Not related" based on the |
| | company's causality assessment provided in "AE matching results" are |
| Adverse reaction | regarded as an adverse reaction. |
| | With adverse reaction: at least 1 record on adverse reaction(s) exists |
| | Without adverse reaction: other than the above. |

| Data name | Derivation and calculation methods |
|---|---|
| | Follow the way of counting adverse events to count adverse reactions. |
| | Based on the seriousness criteria for company assessment which are |
| | provided in "AE matching results", regard the events which have been |
| | assessed to be serious as serious adverse reactions. |
| Serious adverse | With serious adverse reaction: at least 1 record on serious adverse |
| reactions | reaction(s) exists |
| | Without serious adverse reaction: other than the above. |
| | Follow the way of counting adverse events to count serious adverse |
| | reactions. |
| | If more than one identical SOC or PT are found in a patient in counting |
| | adverse events, adverse reactions, serious adverse events, and serious |
| | adverse reactions per outcome, identify the events to be counted with the |
| Outcome | following priority, using the outcomes for company assessment provided |
| | in "AE matching results". |
| | [1] death [2] with sequela [3] not recovered [4] unknown [5] not provided |
| | [6] recovering [7] recovered |
| Death case | At least a piece of data on "death" is found as the outcome of the adverse |
| Death case | events during the safety analysis period. |
| | Use the onset date for company assessment provided in "AE matching |
| | results". |
| | When the first administration date of Humira and the adverse-event onset |
| | date can be identified as the complete date, they can be used for |
| Days from the first | calculation. |
| administration date of | When the first administration date of Humira <= the adverse-event onset |
| Humira to the | date |
| adverse-event onset | Adverse-event onset date - the first administration date of Humira + 1 |
| date | When the first administration date of Humira > the adverse-event onset |
| | date |
| | Adverse-event onset date - the first administration date of Humira |
| | When more than one identical PT is found in a patient, use the first onset |
| | date to identify the adverse event to be counted. |
| Days from the | Use the onset date and the outcome confirmation date (recovered or |
| adverse-event onset | recovering)for company assessment provided in "AE matching results". |
| date to the outcome | When the adverse-event onset date and the outcome confirmation date can |
| confirmation date | be identified as the complete date, they can be used for calculation. |
| (recovered or | Outcome confirmation date - adverse-event onset date + 1 |

| Data name | Derivation and calculation methods |
|---|---|
| recovering) | When more than one identical PT is found in a patient, choose the event which persisted longest until the recovery or the outcome confirmation date. |
| Incidence of adverse reactions, incidence of serious adverse reactions, incidence of adverse events, incidence of serious adverse events | Calculate the incidence of adverse reactions, incidence of serious adverse reactions, incidence of adverse events, incidence of serious adverse events with the number of patients with any of the reactions/events in numerator and the number of patients in the safety analysis group in denominator. Provide how to calculate in each table at Chapter 13 and thereafter if other calculation methods are used. |

## 10.3. Effectiveness analysis

| Data name | Derivation and calculation methods |
|---|---|
| General improvement | Use what has been provided in "general improvement rate (primary |
| rate | physician's assessment" of the survey form. |
| | Partial Mayo score + endoscopic finding score |
| Mayo score | * Only the survey forms with all the scores assessed are calculated (if any |
| | unassessed scores are included, they are excluded from calculation) |
| Remission of Mayo | It should be calculated as 1 or less if the Mayo score is 2 or below and a |
| score | sub-score. |
| | Stool frequency score, rectal bleeding score and physician's global |
| Dontiel Mayo goons | assessment |
| Partial Mayo score | * Only the survey forms with all the scores assessed are calculated (if any |
| | unassessed scores are included, they are excluded from calculation) |
| Remission of partial | It should be calculated as 1 or less if the partial Mayo score is 2 or below |
| Mayo score | and a sub-score. |
| | Partial Mayo score at every assessment decreases by 2 points or more and |
| | by 30% or more in comparison to the partial Mayo score when |
| Improvement of | administration was started. In addition, at least one of the following |
| partial Mayo score | conditions shall be met. |
| (responder) | •Rectal bleeding score has been decreased by at least 1 point since the |
| | administration was started. |
| | • Rectal bleeding score is ≤1. |
| Endoscopy results | Use what has been provided in "endoscopic findings" of the survey form. |

# 11. How to stratify data

| Data | How to stratify |
|---|---|
| Dosage and | 160mg→80mg→40mg once every two weeks and no changes thereafter, |
| administration | other |
| | The first administration to <week (1-28="" 4="" administration,="" days)<="" of="" td=""></week> |
| | ≥Week 4 of administration and <week (29-56="" 8="" administration="" days)<="" of="" td=""></week> |
| | ≥Week 8 of administration and <week (57-168="" 24="" administration="" days)<="" of="" td=""></week> |
| | ≥Week 24 of administration and <week (169-336<="" 48="" administration="" of="" td=""></week> |
| Dose period | days) |
| | ≥Week 48 of administration and ≤Week 52 of administration (337-365 |
| | days) |
| | Unknown |
| | * when the first administration is counted as 1. |
| | ≥1 and ≤4, |
| D | ≥5 and ≤12, |
| Dosing frequency | ≥13 and ≤24, |
| | ≥25 |
| | ≥40mg and ≤500mg, |
| Total dose | ≥501mg and ≤1000mg, |
| | ≥1001mg |
| Reason for | Development of adverse event, lack of effectiveness, patient's wish, no |
| discontinuation | visit, others, multiple answers are acceptable |
| Reason for | Treatment/surgery, pregnancy, concern about the onset of adverse events, |
| discontinuation, other | the condition improved, the condition worsened |
| reasons | Poor adherence, for study |
| Sex | Man, women, unknown/not provided |
| Pregnancy/nursing | Not pregnant/nursing, pregnant, nursing, unknown/not provided |
| Race | Japanese, other Asians, others, unknown/not provided |
| Age (in years) | $<15, \ge 15$ and $<65, \ge 65$ , unknown/not provided |
| | <30, ≥30 and <40, ≥40 and <50, ≥50 and <60, ≥60, unknown/not |
| Body weight (kg) | provided |
| BMI(kg/m <sup>2</sup> ) | $<18.5, \ge 18.5 \text{ and } <25, \ge 25 \text{ and } <30, \ge 30, \text{ unknown}$ |
| Duration of illness (in | |
| years) | $<2, \ge 2$ and $<10, \ge 10$ , unknown/not provided |
| Indication (registration | Colitis ulcerative, others, not provided |
| form) | |

| Data | How to stratify |
|---|---|
| Allergy history | Without the history, with the history, unknown/not provided |
| Smoking history | Without the history, with the history, unknown/not provided |
| Detailed classification of smoking history | Smoking, only in the past (not smoking now), unknown |
| Tuberculosis test | Not conducted, conducted |
| Hepatitis B test | Not conducted, conducted |
| Complications | Without the history, with the history, unknown/not provided |
| Detailed classification of complications | Liver disorder, renal disorder, blood disorder, respiratory disorder, others |
| Other classification of complications | Diabetes mellitus, osteoporosis, malignant tumour, others |
| Medical history | Without the history, with the history, unknown/not provided |
| Detailed classification of medical history | Tuberculosis, non-tuberculous mycobacteriosis, interstitial pneumonia, bronchitis bacterial, aplastic anaemia, pancytopenia, malignant tumour, others |
| Prior medications for colitis ulcerative | Without the history, with the history, unknown/not provided |
| Details classification of | Infliximab, other biological products, aminosalicylic acid products, |
| prior medications for | corticosteroid, azathioprine & 6-mercaptopurine, tacrolimus & |
| colitis ulcerative | ciclosporin, antibiotics, prior medication: others |
| Prior treatment for colitis ulcerative | Without the history, with the history, unknown/not provided |
| Details classification of prior treatment for colitis ulcerative | Leukocytapheresis, surgery, enteral nutrition therapy, intravenous nutrition therapy, others |
| Treatment history with biological products | Without the history, with the history, unknown/not provided |
| Detailed classification of "with" biological products | Infliximab, other biological products Reason for discontinuation: lack of effectiveness Reason for discontinuation: adverse events Reason for discontinuation: others Reason for discontinuation: unknown/not provided |
| Concomitant medications for colitis ulcerative Details classification of | Without the history, with the history, unknown/not provided |
| Details classification of | Aminosalicylic acid products, corticosteroid, azathioprine & |

| Data | How to stratify |
|---|---|
| concomitant | 6-mercaptopurine, tacrolimus & ciclosporin, antibiotics, others |
| medications for colitis | |
| ulcerative | |
| Concomitant therapy | Without the history, with the history, unknown/not provided |
| for colitis ulcerative | without the history, with the history, unknown/hot provided |
| Details classification of | Leukocytapheresis, surgery, enteral nutrition therapy, intravenous |
| concomitant therapy for | nutrition therapy, others |
| colitis ulcerative | nutrition dicrapy, outers |
| Site of disease | Rectum, colon, unknown/not provided |
| Details classification of | |
| a site of disease | Sigmoid, descending, transverse, ascending |
| "colon" | |
| Site of disease by type | Rectal only (no colon), including any of transverse or ascending site, |
| Site of disease by type | others, unknown/not provided |
| Self administration | Without the history, with the history, unknown/not provided |
| Self-administration | Without the history, with the history, unknown/not provided |
| error | without the history, with the history, unknown/hot provided |
| General improvement | Effective or better, ineffective |
| rate | Effective of better, memective |
| Detailed classification | |
| of effective or better of | Markedly effective, effective |
| general improvement | iviairodiy ciicciive, ciicciive |
| rate | |
| Partial Mayo score | $\geq$ 0 and $\leq$ 3, $\geq$ 3 and $\leq$ 6, $\geq$ 6 and $\leq$ 9, unknown/not provided |
| CRP | $<0.3 mg/dL, \ge 0.3 mg/dL$ and $<1 mg/dL, \ge 1 mg/dL$ , unknown/not provided |
| Endoscopy results | normal or remission mucosa, mild, moderate, severe |

## 12. Handling of data for test/assessment periods

## 12.1. Assessment period for the administration status of Humira

Time allowance of assessment period with the first administration date of Humira as 1 is as follows:

| Assessment period | Time Allowance(Day) |
|---|---|
| The first administration to <week 4="" of<="" td=""><td>1~28</td></week> | 1~28 |
| administration | 1~28 |
| ≥Week 4 of administration and <week 8="" of<="" td=""><td>29~56</td></week> | 29~56 |
| administration | 29~30 |
| ≥Week 8 of administration and <week 24="" of<="" td=""><td>57~168</td></week> | 57~168 |
| administration | 3/~108 |
| ≥Week 24 of administration and <week 48="" of<="" td=""><td>169~336</td></week> | 169~336 |
| administration | 109~330 |
| ≥Week 48 of administration and ≤Week 52 of | 337~365 |
| administration | 33/~303 |

## 12.2. Assessment period for the onset status of adverse reactions

Time allowance of assessment period with the first administration date of Humira as 1 is as follows:

| Assessment period | Time Allowance(Day) |
|---|---|
| The first administration to <week 4="" of<="" td=""><td colspan="2" rowspan="2">1-28</td></week> | 1-28 |
| administration | |
| ≥Week 4 of administration and <week 8="" of<="" td=""><td>29-56</td></week> | 29-56 |
| administration | 29-30 |
| ≥Week 8 of administration and <week 24="" of<="" td=""><td>57-168</td></week> | 57-168 |
| administration | 37-168 |
| ≥Week 24 of administration and <week 48="" of<="" td=""><td>169-336</td></week> | 169-336 |
| administration | 109-330 |
| ≥Week 48 of administration and ≤Week 52 of | 337-365 |
| administration | 337-303 |
| > Week 52 of administration | 366- |

#### 12.3. Assessment period for Mayo score

Time allowance of assessment period with the first administration date of Humira as 1 is as follows:

| Assessment period | Time Allowance(Day) |
|---|---|
| At the first administration | -14 ~ 1 (scheduled date: 1) |
| Week 24 of administration | 155 ~ 183 (scheduled date: 169) |
| Week 52 of administration | 337 ~ 393 (scheduled date: 365) |
| A4 diamandian | The final administration date of Humira + 14 (scheduled date: |
| At discontinuation | the final administration date of Humira) |
| At final assessment | Data for the final assessment period among the assessment |
| At imai assessment | applicable to the Time Allowance of each assessment period. |

The data for analysis should derive from the one the closest to the scheduled date within Time Allowance. If there are more than one data dated on the same day, select the higher value.

## 12.4. Assessment period for partial Mayo score

Time allowance of assessment period with the first administration date of Humira as 1 is as follows:

| Assessment period | Time Allowance(Day) |
|---|---|
| At the first administration | -14 ~ 1 (scheduled date: 1) |
| Week 4 of administration | 15 to 42 (scheduled date: 29) |
| Week 8 of administration | 43 to 70 (scheduled date: 57) |
| Week 16 of administration | 98 to 126 (scheduled date: 112) |
| Week 24 of administration | 155 ~ 183 (scheduled date: 169) |
| Week 52 of administration | 337 ~ 393 (scheduled date: 365) |
| At discontinuation | The final administration date of Humira + 14 (scheduled date: |
| | the final administration date of Humira) |
| At final assessment | Data for the final assessment period among the assessment |
| | applicable to the Time Allowance of each assessment period. |

The data for analysis should derive from the one the closest to the scheduled date within Time Allowance. If there are more than one data dated on the same day, select the higher value.

## 12.5. Assessment period for general improvement rate

Time allowance of assessment period with the first administration date of Humira as 1 is as follows:

| Assessment period | Time Allowance(Day) |
|---|---|
| At Week 52 of administration or when the administration is discontinued | Discontinued patients |
| | 1 to the final administration date of Humira + 14 |
| | (scheduled date: the final administration date of Humira) |
| | Other than discontinued patients |
| | 1 to 393 (scheduled date: 365) |

## 12.6. Assessment period for CRP

Time allowance of assessment period with the first administration date of Humira as 1 is as follows:

| Assessment period | Time Allowance(Day) |
|---|---|
| At the first administration | -14 ~ 1 (scheduled date: 1) |
| Week 4 of administration | 15 to 42 (scheduled date: 29) |
| Week 8 of administration | 43 to 70 (scheduled date: 57) |
| Week 24 of administration | 155 ~ 183 (scheduled date: 169) |
| Week 52 of administration | 337 ~ 393 (scheduled date: 365) |
| At discontinuation | The final administration date of Humira + 14 (scheduled date: |
| | the final administration date of Humira) |
| At final assessment | Data for the final assessment period among the assessment |
| At final assessment | applicable to the Time Allowance of each assessment period. |

The data for analysis should derive from the one the closest to the scheduled date within Time Allowance. If there are more than one data dated on the same day, select the higher value.

## 12.7. Assessment period for the continued administration of Humira

The assessment period with the first administration date of Humira as 1 is as follows:

| Assessment period | Day |
|-----------------------------|-----|
| At the first administration | 1 |
| Week 4 of administration | 29 |
| Week 8 of administration | 57 |
| Week 16 of administration | 113 |
| Week 24 of administration | 169 |
| Week 52 of administration | 365 |

## 13. Charts to be generated (chart No., chart name)

## 13.1. General

#### "1.1 Case structure chart"

Patients for analysis: registered patients

Analysis objective: to indicate changes in the number of patients

Analysis items: number of registered sites, number of registered patients, number of sites with patients whose survey form has been locked, number of patients whose survey form was locked, number of patients whose survey form was yet to be locked, number of patients in the safety analysis group, number of patients excluded from the safety analysis group, the breakdown of reasons for exclusion from the safety analysis group, number of patients excluded from the effectiveness analysis group, the breakdown of reasons for exclusion from the effectiveness analysis group

Note: If the reason for exclusion is null for an item, the item itself will not be displayed.

"1.2 The number of sites for survey and the number of patients surveyed"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show the number of patients per site

Analysis items: number of sites with patients whose survey form has been locked, number of patients whose survey form was locked, the mean number of patients per site

To show the maximal, minimal number of patients

"1.3 A list of the patients excluded from the safety analysis group and the patients excluded from the effectiveness analysis group (including the reason for exclusion)"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show the list of patients excluded from each analysis group and the reason for exclusion

Analysis item: The reason for exclusion will not be displayed for the patients not in the safety or efficacy analysis.

If more than one reason for exclusion exists in a patient, display them in a comma-delimited manner.

#### "1.3.1. Excluded patients (aggregation by reason)

Patients for analysis: registered patients

Analysis objective: to show the reason for exclusion in each analysis group regarding all the patients in the analysis group.

Analysis items: patients whose survey form was yet to be locked, patients excluded from the safety analysis group, the breakdown of reasons for exclusion from the safety analysis group, patients

excluded from the effectiveness analysis group, the breakdown of reasons for exclusion from the effectiveness analysis group

Note: After all patients' data are displayed, display "1" at the applicable column. If not applicable, leave the column blank. For "Data credibility not confirmed" in the "reason for exclusion from the safety analysis", display the breakdown. If more than one category for the breakdown exists in a patient, display them in a comma-delimited manner.

"1.4 A list of patients (adverse event + search flag)"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show a list of background information per patient, adverse events and administration status by using analysis data.

Analysis items: case number, sex, age, body weight, duration of illness, adverse event (presence/absence of adverse event, safety

Patients with adverse events not in the analysis period, SOC code, System Organ Class, PT code, name of disease (MedDRA PT), adverse events reported by physician, onset date, days from the first administration to the onset, seriousness, causality, outcome, outcome confirmation date, days to the outcome confirmation), general improvement rate, administration status of Humira (the first administration date, the final administration date, days of administration, the initial dose, the maximum dose), presence/absence of complication, presence/absence of medical history, hepatitis B virus test (HBs antigen, HBs antibody, HBc antibody, HBV-DNA quantitative assay, hepatitis B test), with/without administration of anti-hepatitis B virus agent, tuberculosis (Tuberculin test, QuantiFERON test, T-spot test, chest X ray test, Thoracic CT test, other imaging, tuberculosis test), search flags (patients in the safety analysis group, patients in the effectiveness analysis group, discontinued patients, death cases, pediatrics, the elderly, pregnant, nursing, liver disorder, renal disorder, patients with hepatitis B viral infection, patients with an infection, patients with cytomegalovirus infection, patients with tuberculosis, patients with malignant tumour, patients with administration site reaction, patients with autoimmune disease, patients with pancytopenia, patients with demyelinating disease, patients with cardiac failure congestive, patients with interstitial pneumonia, patients deviated from the administration of Humira, patients with self-administration error, patients with AAA measured, contraindication)

Note: Follow "12.5 Assessment period for general improvement rate" to display the general improvement rate.

Also, display "markedly effective", "effective", "ineffective" and "effectiveness is not assessable". Use 1 (applicable) or 0 (not applicable) to show adverse events which occurred not in the safety analysis period and search flags.

#### "1.4.1 A list of adverse events"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show a list of adverse events per patient by using analysis data.

Analysis items: case number, sex, age, SOC code, System Organ Class, PT code, name of disease (MedDRA PT), adverse events reported by physician, onset date, days from the first administration to the onset, seriousness, causality, outcome, outcome confirmation date, days to the outcome confirmation, complication, patients in the safety analysis group, reason for exclusion from the safety analysis group, patients in the effectiveness analysis group, patients with adverse events not in the safety analysis period, discontinued patients, death cases, pediatrics, the elderly, pregnant, nursing, liver disorder, renal disorder, patients with hepatitis B viral infection, patients with an infection, patients with cytomegalovirus infection, patients with tuberculosis, patients with malignant tumour, patients with administration site reaction, patients with autoimmune disease, patients with pancytopenia, patients with demyelinating disease, patients with cardiac failure congestive, patients with interstitial pneumonia, patients deviated from the administration of Humira, patients with self-administration error, patients with AAA measured, contraindication

Note: The definition of analysis item is the same in "1.4 A list of patients".

Use PT for complications. If a patient has more than one complication, display them in a comma-delimited manner.

### "1.4.2 A list of death cases"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show a list of adverse events in death cases by using analysis data.

Analysis item: Follow "1.4.1 A list of adverse events".

## "1.4.3 A list of prior/concomitant medications in patients with an CMV infection"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show a list of adverse events in patients with an CMV infection by using analysis data.

Analysis item: the patients with at least one PT code in "180111 patients with an CMV infection" among adverse events which occurred in the safety analysis period".

Display the drug name and drug code of prior/concomitant medications for each patient. If more than one drug code exists in a patient, display them in a comma-delimited manner.

## "1.4.4 A list of patients aged 18 years or younger"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show a list of patients aged 18 years or younger by using analysis data.

Analysis items: case number, sex, age, height, body weight, BMI, duration of illness,

discontinued/not discontinued, reason for discontinuation, adverse event (SOC code, System Organ Class, PT code, name of disease (MedDRA PT), onset date, seriousness, causality, outcome, outcome confirmation date), general improvement rate, Administration status of Humira (the first and the final administration dates), complication (PT code, name of disease (MedDRA PT), Medical history (PT code, name of disease (MedDRA PT)), site of disease of colitis ulcerative (rectum, colon, sigmoid, descending, transverse, ascending), Mayo score (at the first administration, Week 24 and Week 52 of administration), Partial Mayo score (at the first administration, Week 8, Week 24, and Week 52 of administration), Search flag (prior medication (Infliximab, other biological products, aminosalicylic acid drug, corticosteroids, azathioprine & 6-mercaptopurine, tacrolimus & ciclosporin, antibiotics))

### "1.5 Administration status of Humira (dosage and administration)"

Patients for analysis: patients in the safety analysis group, patients in the effectiveness analysis group

Analysis objective: to show the administration status of Humira

Analysis items: calculate the number of patients in the analysis groups as well as the percentage to the number of patients and the number of those in the analysis groups per segment defined in "administration status (dosage and administration)" of "10.1 General".

#### "1.5.1 other dosage and administration (a list)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show a list of reasons for change in dose/dosing frequency in patients classified into the dose and administration "others".

Analysis items: Select the patients who are categorized in "others" defined in "administration status (dose and administration)" of "10.1 General", and display the case number and the reason for the change in dose/dosing frequency.

If more than one reason exists in a patient, display them in a comma-delimited manner.

Note: Follow the definition in "the reason for the change in dose/dosing frequency" of "10.1 General" for the reason for the change in dose/dosing frequency.

#### "1.6 Administration status of Humira (dosing frequency, dose)

Patients for analysis: patients in the safety analysis group, patients in the effectiveness analysis group

Analysis objective: to show the dosing frequency and the distribution status of the total dose

Analysis items: calculate the number of patients per segment defined in "11 How to stratify data" as well as the percentage to the number of patients in the analysis groups regarding dosing frequency and the total dose. In addition, calculate summary statistics for each measurement.

#### "1.6.1 Administration status of Humira (period)"

Patients for analysis: patients in the safety analysis group, patients in the effectiveness analysis group

Analysis objective: to show the distribution status in the administration period.

Analysis item: Calculate the administration dates based on "days to the final administration date of Humira" of "10.1 General" as well as the number of patients in the analysis groups. Then, calculate the number of patients per segment which contains the administrations date in each patient and the percentage to the patients in the analysis group in the Time Allowance defined in "12.1 Assessment period for administration status of Humira" In addition, calculate summary statistics for the number of days for administration.

#### "1.6.2 Continuation rate of Humira"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the continuation rate of Humira using the Kaplan-Meier method.

Analysis items: At Risk, number of discontinued patients, continuation rate (the percentage to the number of discontinued patients for At Risk), 95% of continuation rate

Calculate the confidence interval by assessment period. In addition, generate the Kaplan-Meier curve for the continuation rate.

Note: Follow "12.7 Assessment period for the continuation of Humira administration" for the dates of assessment period.

The days are censored at the first administration date of Humira + 364 in patients who are still registered at Week 52.

Calculate the analysis items using the Kaplan-Meier method.

At Risk should include the number of patients who are exposed to a discontinuation risk.

#### "1.7 Administration status of Humira (discontinuation of administration)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the number of discontinued patients and the breakdown of the reasons for discontinuation.

Analysis items: Calculate the number of patients in the analysis groups, the percentage to the discontinued patients and patients in the analysis groups, patients 'with' reason for discontinuation and unknown/not provided and the percentage to the number of discontinued patients, number of patients per "reason for discontinuation" defined in "11 How to stratify data" and the percentage to the number of discontinued patients.

Note: the reasons for discontinuation may be overlapped in calculation.

In addition, if there are no patients applicable to "multiple choices", do not display it per item.

#### "1.7.1 Administration status of Humira (reason for discontinuation other reasons)

Patients for analysis: patients in the safety analysis group

Analysis objective: to show a list in which the reason for discontinuation is others'.

Analysis item: Calculate the number of patients classified into "others " of "reasons for discontinuation" defined in "11 How to stratify data" by segment of "reason for discontinuation, other reason". Display the segments in descending order of number of patients.

#### "1.12 Distribution status of patient backgrounds"

Patients for analysis: patients in the safety analysis group, patients in the effectiveness analysis group, patients whose survey form was locked

Analysis objective: to show the distribution status of patient backgrounds

Analysis item: calculate the number of patients in the analysis groups.

Calculate the number of patients per the following segment defined in "11 How to stratify data" and the percentage to the number of patients in the analysis groups. In addition, calculate summary statistics for each measurement.

Sex, pregnancy/nursing, race, age (year), body weight (kg), BMI (kg/m²), duration of illness (year), indication (registration form), allergy history, smoking history, detailed classification of smoking history, tuberculosis test, hepatitis B test, complication, detailed classification of complications, complication/others, medical history, detailed classification of medical history, prior medication for colitis ulcerative, detailed classification of prior medication for colitis ulcerative, treatment for colitis ulcerative, detailed classification of medical product, concomitant medication for colitis ulcerative, detailed classification of "with" biological product, concomitant medication for colitis ulcerative, detailed classification of concomitant medication for colitis ulcerative, concomitant treatment for colitis ulcerative, detailed classification of the disease site "colon", site of disease by type, partial Mayo score, CRP

Note: For the discontinuation reasons for the detailed classification of pregnant/nursing or 'using' biological products", calculate the percentage to the aggregation item right above the item. For other items, calculate the percentage to the number of target patients.

Overlapped aggregation may occur in the detailed classification of complications and complication of other classification, detailed classification of medical history, detailed classification of prior medications for colitis ulcerative, detailed classification of prior treatment for colitis ulcerative, detailed classification of concomitant medications for colitis ulcerative, detailed classification of concomitant treatment for colitis ulcerative, and the detailed classification of site of disease for colitis ulcerative and the site of

disease "colon".

"1.13 Incidence of self-administration error"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the distribution status for presence/absence of self-administration and the detailed classification of self-administration.

Analysis item: calculate the number of patients in the analysis groups.

Calculate the number of patients per "self-administration" defined in "11. How to stratify data" and the percentage to the number of patients in the analysis groups.

In addition, calculate the number of patients per "self-administration error" and the percentage to the patients 'with' self-administration.

### "1.16 A list of patients with AAA measured

Patients for analysis: patients in the safety analysis group

Analysis objective: to show a list of patients with AAA measured.

Analysis item: display the following items in "patients with AAA measured" defined in "10.1 General".

Case number, administration status of Humira (the first and final administration dates), concomitant medications, serum anti-adalimumab antibody (blood sampling date, positive/negative) adverse events reported by physician, name of disease (MedDRA PT), System Organ Class, onset date, seriousness, causality, outcome confirmation date, outcome, general improvement rate

Note: Show "continued" for patients who are still registered in the survey.

Obtain information on serum anti-adalimumab antibody from "UC Survey AAA Measurement (periodic safety report).

Follow "12.5 Assessment period for general improvement rate" for the general improvement rate.

#### 13.2. Safety

"2.1 A list of onset status of adverse reactions/infections (Attachment Form 2)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of adverse reactions

Analysis item: aggregate the following items by period for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of sites surveyed, number of patients surveyed, number of patients with adverse reactions, etc. number of adverse reactions, incidence of adverse reactions, etc., and type of adverse reactions, etc. (SOC, PT).

Note: the classification of the period is as follows:

The 6th periodic safety report: at approval, from June 14, 2013 to December 31, 2015, from January 1, 2016 to December 31, 2016, cumulative, total

Re-examination: at approval, June 14, 2013 to December 31, 2015, January 1, 2016 to December 31, 2016, January 1, 2017 to May 15, 2017, cumulative, total.

Final report: at approval, cumulative, total

Put \* before the PT of unexpected events from "Precautions".

"2.1.1 A list of the onset status of adverse reactions/infections (patients not in the safety analysis)"

Patients for analysis: patients excluded from the safety analysis group

Analysis objective: to show the onset status of adverse reactions, etc. in patients not in the safety analysis group.

Analysis item: aggregate the following items for adverse reactions which occurred in the safety analysis period:

Calculate the number of patients and the percentage to the number of patients surveyed per number of sites surveyed, number of patients surveyed, number of patients with adverse reactions, etc. number of adverse reactions, incidence of adverse reactions, etc., and type of adverse reactions, etc. (SOC, PT).

"2.1.2 A list of the onset status of adverse reactions/infections not in the follow-up period"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show the onset status of adverse reactions, etc. which occurred not in the follow-up period.

Analysis item: aggregate the following items for adverse reactions which occurred not in the safety analysis period:

Calculate the number of patients and the percentage to the number of patients surveyed per number of sites surveyed, number of patients surveyed, number of patients with adverse reactions, etc. number of adverse reactions, incidence of adverse reactions, etc., and type of adverse reactions, etc. (SOC, PT).

"2.2 A list of the onset status of serious adverse events (Attachment Form 10)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of serious adverse events

Analysis item: aggregate the following items per period for adverse events which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number

of sites surveyed, number of patients surveyed, number of patients with serious adverse events, number of serious adverse events, incidence of adverse events, incidence of serious adverse events and type of adverse reactions, etc. (SOC, PT).

Note: see "2.1 A list of the onset status of adverse reactions/infections (Attachment Form 2)" on how to separate the period.

Put \* before the PT of unexpected events from "Precautions".

#### "2.3 A list of target-patient summary (Attachment Form 3)"

Patients for analysis: patients whose survey form was locked

Analysis objective: to show a list of patients

Analysis item: provide the items for analysis and the definitions below.

(1) Case number

Provide a serial number starting 1 per patient.

(2) Name of site (company code)

Describe it in Japanese, as the official name. Obtain the name of site from "[Humira UC]DCF code list Company A" and "[Humira UC]DCF code list Company E".

(3) Main establishing entity/code

Obtain the code from "Ultmarc re-examination classification".

(4) Name of prefecture where the business is located

Fill in the name. Obtain the prefecture's name from "Ultmarc re-examination classification".

(5) Patient abbreviation name

Fill in "not applicable" as mentioned in GB.

(6) Sex

Fill in man, women, unknown or not provided as mentioned in GB.

(7) Date of birth (or age)

Unify it in age. Fill in "A + age + "0000" as mentioned in GB.

(8) Inpatient/outpatient

Fill in inpatient, outpatient, unknown or not provided as mentioned in GB.

(9) Indication

Code, name of disease: Obtain the MedDRA/J PT code and PT from the indication of Humira described in the survey form. If the indication is 'other', obtain the indication from "[Humira UC] indication, other detailed coding".

(10) Severity prior to administration

Four stages of "physician's global assessment" at first administration in "Effectiveness assessment (partial Mayo-score)" of the survey form: remission phase, mild, moderate and severe

Select the data dated before the first administration date. If the date is behind the first administration date, select "no assessment". If the date is not provided or unknown, select

"unknown".

#### (11) Complications

Presence/absence: Refer to the "presence/absence of complications" defined in "10.1 General".

Number of described complications: the number of PT codes encoded by MedDRA/J. If more than 1 identical PT code is found in a patient, count the PT as 1. Describe "0" for the case with no complications.

Term: Describe the PT of complication encoded by MedDRA/J. Arrange detailed classification of complication, the name of complication disease name, a serial number of the complication per patient. Leave the column blank for the case with no descriptions.

#### (12) Route of administration

Describe it as "SC".

#### (13) Maximal dose (a day/volume)

The daily maximum dose Select the largest number in "administration status (dose and administration) defined in "10.1 General" per patient.

## (14) The mean dose (a day/volume)

The mean daily dose

It should be the value of "total dose/total dosing times" based on the "administration status (total dosing time, total dose)" defined in "10.1 General".

#### (15) Unit

Use "MG".

### (16) daily dosing frequency (the maximum)

Use "1".

#### (17) Period for administration

The value of "total dosing time" based on "administration status (total dosing time, total dose)" defined in "10.1 General".

#### (18) Concomitant medications

Drug code, the principal drug name: arrange them with sequence with the priority of concomitant medications for colitis ulcerative per patient, and choose the top concomitant medication. If there is no concomitant medication, leave the drug code column blank, and the name of the primary drug "null".

Number of descriptions: count the number of drug codes arranged as mentioned above. If more than 1 identical drug code is found in a patient, count it as 1. Describe "0" for the case with no concomitant medications.

#### (19) Effectiveness level

Display the general improvement rate calculated in accordance with "12.5 Assessment period of general improvement rate". Of note, as for the patients with no general improvement rate calculated in accordance with 12.5, if there is a description on the assessment in the survey form, use the description. If not, display "not described". If it is not assessable, display "unknown".

#### (20) Adverse reactions

Handle the events with the identical PT code in a patient as 1 record regarding adverse events which occurred in the safety analysis period.

Organ-name code: select the SOC code. When presence/absence is "absence", leave the column blank.

Adverse reaction code: select the PT code. When presence/absence is "absence", leave the column blank.

Name of adverse reactions: select the PT. When presence/absence is "absence", leave the column blank.

Presence/absence: Select "present" for the data with both adverse events and causal relationship among the adverse reactions which occurred in the safety analysis period. If presence/absence of adverse events is unknown, select "unknown". If presence/absence of adverse events is not provided, select "not provided". Others are "absent". If the reason is 'safety assessment cannot be made' in the patients excluded from the safety analysis, select "unknown".

Number of descriptions: count the number of PT codes. If more than 1 identical PT code is found in a patient, count the PT as 1.

When presence/absence is "absence", leave the column blank.

#### (21) Outcome

For PT codes displayed for adverse reactions, select the outcome with the highest priority in the "outcome" priorities defined in "10.2 Safety analysis". When presence/absence of adverse reactions is "absence", leave the column blank.

#### (22) Survey form number

Use the case number in this study.

#### (23) Dropout

If a patient is dropped out from both the safety analysis and the effectiveness analysis, display the case as "both dropout".

If a patient is dropped out only from the safety analysis, display the case as "Safe dropout".

"If a patient is dropped out only from the effective analysis, display the case as "Effective\_dropout".

Note: If there are no applicable data in an aggregation column, display "0" and no columns should be left blank.

#### "2.4.1 A list of the onset status of adverse reactions (priority survey items)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the summary statistics on the days to the onset as well as the number of patients per outcome and the days to the confirmed outcome (recovered or recovering) for adverse reactions of the priority survey items.

Analysis items: calculate the number of cases and the percentage to the number of patients in the analysis groups per type of adverse reactions (priority survey item, PT), and the number of patients with serious reactions and the percentage to the number of patients in the analysis groups regarding the adverse reactions which occurred in the safety analysis period. In addition, calculate the summary statistics (the number of patients, the mean, the minimum, the median, the maximum) for days to the onset per PT and priority survey item (for the total number of PTs) and for days from the onset date to the outcome (recovered or recovering) as well as the number of patients per outcome.

Note: When more than one identical PT is found in a patient, aggregate seriousness, days to the onset, outcome and days to the outcome (recovered or recovering) as 1 patient (case) in the following manner.

- Seriousness priority: serious > non-serious
- Days to the onset: identify the days as mentioned in "days from the first administration date of Humira to the adverse-event onset date" defined in "10.2 Safety analysis".
- Outcome: identify it as mentioned in "outcome" defined in "10.2 Safety analysis".
- Days to outcome (recovered or recovering): identify the days as mentioned in "days from the first administration date of Humira to the outcome confirmation date (recovered or recovering)" defined in "10.2 Safety analysis".

"2.4.2 A list of the onset status of adverse reactions (identified important risks)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the summary statistics of the days to the onset, the number of patients per outcome, and the days to the onset and the days to the outcome (recovered or recovering) regarding the adverse reactions of identified important risks based on "20180115\_how to extract risks (RMP)\_MedDRA20.1".

Analysis items: calculate the number of cases and the percentage to the number of patients in the analysis groups and the number of patients with serious reactions and the percentage to the number of patients in the analysis groups per type of identified important risks (identified important risks, PT), regarding the adverse reactions which occurred in the safety analysis period. In addition, calculate the summary statistics (the number of patients, the mean, the minimum, the median, the maximum) for days to the onset per PT and identified important risks (the total number of PTs) and for days from the onset date to the outcome (recovered or recovering) as well as the number of patients per outcome.

Note: When more than one identical PT is found in a patient, refer to "2.4.1 A list of the onset status of adverse reactions (priority survey items)"

#### "2.4.3 A list of the onset status of adverse events (priority survey items)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the summary statistics on the days to the onset as well as the number of patients per outcome and the days to the confirmed outcome (recovered or recovering) for adverse events of the priority survey items.

Analysis item: handle the items for analysis and definitions as mentioned in "2.4.1 A list of the onset status of adverse reactions (priority survey item)" for adverse events which occurred in the safety analysis period.

#### "2.4.4 A list of the onset status of adverse events (identified important risks)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the summary statistics of the days to the onset, the number of patients per outcome, and the days to the onset and the days to the outcome (recovered or recovering) regarding the adverse events of identified important risks based on "20180115\_how to extract risks (RMP) MedDRA20.1".

Analysis item: handle the items for analysis and definitions as mentioned in "2.4.2 A list of the onset status of adverse reactions (identified important risks)" for adverse events which occurred in the safety analysis period.

#### "2.5 A list of the onset status of adverse reactions with/without self-administration"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of adverse reactions with/without self-administration Analysis item: aggregate the following items with/without self-administration for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, etc. number of adverse reactions, type of adverse reactions, etc. (SOC, PT).

#### "2.5.1 A list of the onset status of adverse reactions with/without self-administration"

Patients for analysis: patients excluded from the safety analysis group

Analysis objective: to show the onset status of adverse reactions with/without self-administration Analysis item: aggregate the following items with/without self-administration for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, etc. number of adverse reactions, type of adverse reactions, etc. (SOC, PT).

"2.6 Incidence of adverse reactions per onset period (serious)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of serious adverse reactions per the onset period.

Analysis item: aggregate the following items by period for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with serious adverse reactions, etc. type of adverse reactions, etc. (SOC, PT).

Note: Aggregate the initial events among the identical PTs in a patient. Aggregate the events based on the segments which contain the initial onset period of adverse reactions among Time Allowance defined in "12.2 Assessment period for the onset status of adverse reactions". When calculating the number of patients with the target events, remove unnecessary data per case number and onset period. When calculating the number of SOC, remove unnecessary data per case number, onset period and SOC.

Count the number of patients surveyed by using the date defined below until the assessment period applicable to Time Allowance defined in "12.2 Assessment period for the onset status of adverse reactions".

- Discontinued patients: the final administration date of Humira + 28 days
- Not discontinued patients: the first administration date of Humira + 392 days

Even if there is one adverse reaction, it should be counted as one patient in every period when the reaction persisted.

"2.7 Incidence of adverse reactions per set period"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of adverse reactions per onset period.

Analysis item: aggregate the following items by period for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, etc. type of adverse reactions, etc. (SOC, PT).

Note: Refer to the note of "2.6 Incidence of adverse reactions per onset period (serious)".

"2.9 Incidence of adverse reactions (serious adverse reactions/adverse reactions) per background factor"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the incidence of adverse reactions per patient background factor and

analyze them.

Analysis items: calculate the number of all patients, the percentage to the number of patients with serious adverse reactions and all patients, the number of patients with adverse reactions and the percentage to number of all patients, the tests for adverse reactions (Fisher's exact test for nominal-scale factors and Man-Whitney's u test for ordinal-scale factors) per the following patient background factor regarding the adverse reactions which occurred in the safety analysis period.

Note: the patient background factors are as follows:

Age (year), the elderly, pediatrics, sex, body weight (kg), BMI (kg/m<sup>2</sup>), duration of illness (year), complications, complication: hepatic function disorder, complication; renal impairment, complication: blood disorder, complication: respiratory disorder, complication: diabetes mellitus, complication: osteoporosis, complication: malignant tumour, medical history, medical history: tuberculosis, medical history: non-tuberculous mycobacteriosis, medical history: interstitial pneumonia, medical history: bronchitis bacterial, medical history: aplastic anaemia, medical history: pancytopenia, medical history: malignant tumour, allergy history, smoking history, detailed history of smoking history, the administration status of Humira: self-administration, prior medication, prior medication: biological product, prior medication Infliximab, prior medication: other biological product, prior medication: aminosalicylic acid drug, prior medication: corticosteroids, prior medication: azathioprine, prior medication 6-mercaptopurine, prior medication: azathioprine & 6-mercaptopurine, prior medication: tacrolimus & ciclosporin, prior treatment, prior treatment: leukocytapheresis, prior treatment: surgery, prior treatment: enteral nutrition therapy, prior treatment: intravenous nutrition therapy, concomitant medication, concomitant medication: aminosalicylic acid drug, concomitant medication: corticosteroids, concomitant medication: azathioprine, concomitant medication: 6-mercaptopurine, concomitant medication: azathioprine & 6-mercaptopurine, concomitant medication: tacrolimus & ciclosporin, concomitant treatment, concomitant treatment: leukocytapheresis, concomitant treatment: surgery, concomitant treatment: intravenous nutrition therapy, concomitant treatment: enteral nutrition therapy, site of disease by type, partial Mayo score, **CRP** 

"2.9.xx Incidence of adverse reactions per background factor and seriousness"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of non-serious/serious adverse reactions per statistically-significant background factor based on the test results in 2.9.

Analysis item: aggregate the following items per background factor and seriousness for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, incidence of the reactions, number of adverse reactions and type of adverse reactions (SOC, PT).

"2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of non-serious/serious adverse reactions with/without hepatic function disorder

Analysis item: aggregate the following items with/without hepatic function disorder per seriousness regarding the adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, incidence of the reactions, number of adverse reactions and type of adverse reactions (SOC, PT).

Note: Aggregate the most serious reaction among the identical PTs in a patient.

When calculating the number of patients with the target events, remove unnecessary data per case number and seriousness. When calculating the number of SOC, remove unnecessary data per case number, seriousness and SOC.

"2.14.1 Incidence of adverse reactions with/without renal impairment and per seriousness" Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of non-serious/serious adverse reactions with/without renal impairment

Analysis items: aggregate the following items with/without renal impairment per seriousness regarding the adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, incidence of the reactions, number of adverse reactions and type of adverse reactions (SOC, PT).

Note: refer to the note of "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness".

"2.15.1 Incidence of adverse reactions per seriousness in pediatrics and non-pediatrics"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of adverse reactions in pediatrics and non-pediatrics per outcome.

Analysis items: aggregate the following items per seriousness in pediatrics and non-pediatrics regarding adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, incidence of the reactions, number

of adverse reactions and type of adverse reactions (SOC, PT).

Note: refer to the note of "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness".

"2.16.1 Incidence of adverse reactions per seriousness in the elderly and non-elderly patients" Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of non-serious/serious adverse reactions in the elderly and non-elderly patients.

Analysis items: aggregate the following items per seriousness in the elderly and non-elderly patients regarding adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, incidence of the reactions, number of adverse reactions and type of adverse reactions (SOC, PT).

Note: refer to the note of "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness".

"2.17 A list of the onset status of adverse reactions/infections in this survey"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of adverse reactions, etc. and serious adverse reactions, etc.

Analysis item: aggregate adverse reactions and serious adverse reactions regarding the following items based on the adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, etc. number of adverse reactions, incidence of adverse reactions, etc., and type of adverse reactions, etc. (SOC, PT).

Note: refer to the note of "2.13.1 Incidence of adverse reactions with/without hepatic function disorder and per seriousness" for serious adverse reactions.

"2.18 A list of the onset status of adverse reactions with/without treatment history with biological products".

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of adverse reactions with/without treatment history with biological products.

Analysis item: aggregate the following items with/without treatment history with biological products for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, incidence of the reactions, number of adverse reactions and type of adverse reactions (SOC, PT).

"2.18.1 A list of the onset status with/without treatment history with biological products (patients excluded from the safety analysis group)"

Patients for analysis: patients excluded from the safety analysis group

Analysis objective: to show the onset status of adverse reactions with/without treatment history with biological products.

Analysis item: aggregate the following items with/without treatment history with biological products for adverse reactions which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, incidence of the reactions, number of adverse reactions and type of adverse reactions (SOC, PT).

#### "2.19 A list of the onset status of adverse events in this survey"

Patients for analysis: patients in the safety analysis group

Analysis objective: to show the onset status of adverse events, serious adverse events and non-serious adverse events.

Analysis items: aggregate adverse events, serious adverse events and non-serious adverse events regarding the following items among adverse events which occurred in the safety analysis period.

Calculate the number of patients and the percentage to the number of patients surveyed per number of patients surveyed, number of patients with adverse reactions, number of adverse reactions, incidence of the reactions, type of adverse events (SOC, PT).

Note: When more than one identical PT is found in a patient, aggregate the event as 1 patient (case) in the following manner:

• Seriousness priority: serious > non-serious

#### "2.20 A list of the onset status of adverse reactions (all cases)"

Patients for analysis: patients in the safety analysis group

Analysis objective: to calculate the following items by seriousness for adverse reactions which occurred in the safety analysis period. Calculate the number of patients and the percentage to the number of patients surveyed per number of patients with adverse reactions, incidence of the reactions, number of adverse reactions and type of adverse reactions (SOC, PT). In addition, show the number of cases per days to outcome (recovered or recovering), number of patients per outcome, summary statistics of days to the onset per type of adverse reactions (PT).

Note: When more than one identical PT is found in a patient, aggregate seriousness, days to the onset, outcome and days to the outcome (recovered or recovering) as 1 patient (case) in the following manner.

• Seriousness priority: serious > non-serious

• Days to the onset: identify the days as mentioned in "days from the first administration date of Humira to the adverse-event onset date" defined in "10.2 Safety analysis".

• Outcome: identify it as mentioned in "outcome" defined in "10.2 Safety analysis".

 Days to outcome (recovered or recovering): identify the days as mentioned in "days from the first administration date of Humira to the outcome confirmation date (recovered or recovering)" defined in "10.2 Safety analysis".

#### 13.3. Effectiveness

"3.1.1 Changes in Mayo score (Observed Case)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show Mayo score and the changes in Mayo score per assessment period.

Analysis item: calculate the number of patients in the analysis groups.

Calculate the number of target patients, the mean and standard deviation of Mayo score, the mean and standard deviation of changes in Mayo score for each assessment period, and conduct a paired-t test which compares the values at the initial administration.

Note: Follow "12.3 Assessment period for Mayo score" for Time Allowance of assessment period.

The analysis covers only the patients with the assessment applicable to Time Allowance of the first administration and each assessment period.

Multiplicity in the test will be adjusted by the Bonferroni method.

"3.1.2 Changes in the remission rate at each point of Mayo score (Observed Case)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show the remission rate of Mayo score per assessment period.

Analysis item: calculate the number of patients in the analysis groups.

Calculate the number of target patients, the percentage to the number of patients who achieved a remission and the number of target patients, 95%CI of the remission rate, and conduct a McNemar test for the first administration per assessment period.

In addition, prepare a line plot to describe the percentage to the target patients among the patients who achieved a remission per assessment period.

X-axis: assessment period (in week)

Y-axis: percentage (%)

Note: Follow "12.3 Assessment period for Mayo score" for Time Allowance of assessment period.

The analysis covers only the patients with the assessment applicable to Time Allowance of the first administration and each assessment period.

For the confidence interval, use the Clopper-Pearson's confidence interval.

Refer to "10.3 Effectiveness analysis" for the calculation method and remission rate.

#### "3.1.4 Changes in partial Mayo score (Observed Case)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show partial Mayo score and the changes in partial Mayo score per assessment period.

Analysis item: calculate the number of patients in the analysis groups.

Calculate the number of target patients, the mean and standard deviation of partial Mayo score, the mean and standard deviation of changes in partial Mayo score for each assessment period, and conduct a paired-t test which compares the values at the initial administration.

In addition, calculate the mean of the mean days to the final assessment and the standard deviation.

Note: Follow "12.4 Assessment period for partial Mayo score" for Time Allowance of assessment period.

The analysis covers only the patients with the assessment applicable to Time Allowance of the first administration and each assessment period.

Multiplicity in the test will be adjusted by the Bonferroni method.

#### "3.1.5.1 Changes in the remission rate at each point of partial Mayo Score (Observed Case)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show the remission rate of partial Mayo score per assessment period.

Analysis item: calculate the number of patients in the analysis groups.

Calculate the number of target patients, the percentage to the number of patients who achieved a remission and the number of target patients, 95%CI of the remission rate, and conduct a McNemar test for the first administration per assessment period.

In addition, prepare a line plot to describe the percentage to the target patients among the patients who achieved a remission per assessment period.

X-axis: assessment period (in week)

Y-axis: remission rate (%)

Note: Follow "12.4 Assessment period for partial Mayo score" for Time Allowance of assessment period.

The analysis covers only the patients with the assessment applicable to Time Allowance of the first administration and each assessment period.

For the confidence interval, use the Clopper-Pearson's confidence interval.

Refer to "10.3 Effectiveness analysis" for the calculation method and remission rate.

"3.1.5.2 Changes in the remission rate (NRI) at each point of partial Mayo Score"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show the remission rate of partial Mayo score per assessment period.

Analysis item: calculate the number of patients in the analysis groups.

Calculate the number of target patients, the percentage to the number of patients who achieved a remission and the number of target patients, 95%CI of the remission rate, and conduct a McNemar test for the first administration per assessment period.

In addition, prepare a line plot to describe the percentage to the target patients among the patients who achieved a remission per assessment period.

X-axis: assessment period (in week)

Y-axis: remission rate (%)

Note: Follow "12.4 Assessment period for partial Mayo score" for Time Allowance of assessment period.

The analysis covers only the patients with the assessment applicable to Time Allowance of the first administration and each assessment period.

For the confidence interval, use the Clopper-Pearson's confidence interval.

Refer to "10.3 Effectiveness analysis" for the calculation method and remission rate.

NRI: when it is unknown whether the remission is achieved, impute the data without remission.

"3.1.7.1 Remission rate at Week 52 in patients who achieved a remission at Week 8 of administration based on partial Mayo score"

Patients for analysis: Patients in the effectiveness analysis group (the patients who did not achieve a remission when the administration was started but achieved the remission at Week 8 of administration in partial Mayo score)

Analysis objective: to show the remission rate of partial Mayo score at Week 52 of administration in patients in the analysis group.

Analysis items: calculate the number of target patients, the percentage to the number of patients who achieved a remission at Week 52 of administration and the target patients, and the confidence interval of the remission rate. (calculate them in both Observed Case and NRI patterns)

Note: the patients for analysis should have partial Mayo score at the first administration and Week 8 of administration and achieved a remission at Week 8 of administration except those who had already achieved a remission in partial Mayo score at the first administration.

Follow "12.4 Assessment period for partial Mayo score" for Time Allowance of assessment period.

For the confidence interval, use the Clopper-Pearson's confidence interval.

"3.1.7.2 Remission rate at Week 52 in patients who achieved the response as an index of partial Mayo score at Week 8 of administration"

Patients for analysis: Patients in the effectiveness analysis group (the patients who achieved a response at Week 8 of administration in partial Mayo score)

Analysis objective: to show the remission rate of partial Mayo score at Week 52 of administration in patients in the analysis group.

Analysis items: calculate the number of target patients, the percentage to the number of patients who achieved a remission at Week 52 of administration and the target patients, and the confidence interval of the remission rate. (calculate them in both Observed Case and NRI patterns)

Note: the patients for analysis should have partial Mayo score at the first administration and Week 8 of administration and be a responder at Week 8 of administration.

Follow "12.4 Assessment period for partial Mayo score" for Time Allowance of assessment period. For the confidence interval, use the Clopper-Pearson's confidence interval.

Definition of responder: partial Mayo score at every assessment decreases by 2 points or more and by 30% or more. In addition, at least one of the following conditions shall be met.

- Rectal bleeding score has been decreased by at least 1 point since the administration was started.
- Rectal bleeding score is  $\leq 1$ .

#### "3.2 General improvement rate"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show the general improvement rate at Week 52 or at discontinuation of administration

Analysis item: calculate the number of patients in the analysis groups.

For the general improvement rate at the final observation which was calculated according to "12.5 Assessment period of general improvement rate", calculate the percentage to the number of patients and the patients in the analysis group per "general improvement rate" and "detailed classification for patients with an effective or better result in general improvement rate" defined in "11 How to stratify data".

"3.4 Aggregation for effectiveness per patient background factor (general improvement rate)" Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show the effectiveness rate of the general improvement rate at Week 52 or at discontinuation of administration as the primary endpoint and analyze the factors.

Analysis items: calculate the number of patients, the percentage to the number of patients with an effective (markedly effective + effective) in general improvement rate and all patients, the

percentage to the number of patients with an ineffective result in general improvement rate and the number of all patients, the tests for effectiveness (Fisher's exact test for nominal-scale factors and Man-Whitney's u test for ordinal-scale factors) per the following patient background factor.

Note: the patient background factors are as follows:

Age (year), the elderly, pediatrics, sex, body weight (kg), BMI (kg/m<sup>2</sup>), duration of illness (year), complications, complication: hepatic function disorder, complication; renal impairment, complication: blood disorder, complication: respiratory disorder, complication: diabetes mellitus, complication: osteoporosis, complication: malignant tumour, medical history; medical history: tuberculosis, medical history: non-tuberculous mycobacteriosis, medical history: interstitial pneumonia, medical history: bronchitis bacterial, medical history: aplastic anaemia, medical history: pancytopenia, medical history: malignant tumour, allergy history, smoking history, detailed history of smoking history, the administration status of Humira: self-administration, prior medication, prior medication: biological product, prior medication Infliximab, prior medication: other biological product, prior medication: aminosalicylic acid drug, prior medication: corticosteroids, prior medication: azathioprine, prior medication 6-mercaptopurine, prior medication: azathioprine & 6-mercaptopurine, prior medication: tacrolimus & ciclosporin, prior treatment, prior treatment: leukocytapheresis, prior treatment: surgery, prior treatment: enteral nutrition therapy, prior treatment: intravenous nutrition therapy, concomitant medication, concomitant medication: aminosalicylic acid drug, concomitant medication: corticosteroids, concomitant medication: azathioprine, concomitant medication: 6-mercaptopurine, concomitant medication: azathioprine & 6-mercaptopurine, concomitant medication: tacrolimus & ciclosporin, concomitant treatment, concomitant treatment: leukocytapheresis, concomitant treatment: surgery, concomitant treatment: intravenous nutrition therapy, concomitant treatment: enteral nutrition therapy, site of disease by type, partial Mayo score, CRP

## "3.4.1 Aggregation for effectiveness per patient background factor (partial Mayo score)" Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show the remission of partial Mayo score at the final assessment as the primary endpoint per patient background factor and analyze them.

Analysis items: calculate the number of all patients, the percentage to the number of patients who achieved a remission in partial Mayo score and all patients, the number of patients who failed to achieve a remission in partial Mayo score and the percentage to number of all patients, the tests for remission (Fisher's exact test for nominal-scale factors and Man-Whitney's u test for ordinal-scale factors) per the following patient background factor:

Note: Refer to "3.4 Aggregation for effectiveness per patient background factor (general improvement rate)" for patient background factors.

#### "3.5 Changes in CPR level"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show measured CPR levels at each assessment period.

Analysis items: calculate CRP's summary statistics (number of cases, mean, standard deviation, minimum value, 1st quartile value, the median, 3rd quartile value and the maximum value) per assessment period.

Note: Follow "12.6 Assessment period for CRP" for Time Allowance of assessment period.

The analysis covers only the patients with the assessment applicable to Time Allowance of the first administration and each assessment period.

"3.6 The status of corticosteroid use and the remission in partial Mayo score in patients who used corticosteroids when administration was started (Observed Case)"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show the status of corticosteroid use and with/without remission in partial Mayo score per assessment period in patients who concomitantly used corticosteroids when administration was started

Analysis items: calculate the number of target patients, the percentage to the number of patients with/without concomitant use of corticosteroids and to the number of target patients, and the percentage to the number of patients who achieved/failed to achieve a remission in partial Mayo score and to the number of target patients.

Note: The target patients to be counted in each assessment period shall receive Humira in each Time Allowance defined in "12.4 Assessment period of partial Mayo score".

The target patients who concomitantly used corticosteroids at each assessment period shall receive corticosteroids at each scheduled date defined in "12.4 Assessment period of partial Mayo score".

Follow "12.4 Assessment period for partial Mayo score" for Time Allowance of the assessment period regarding with/without remission in partial Mayo score.

## "3.7 Endoscopy results during administration period"

Patients for analysis: patients in the effectiveness analysis group

Analysis objective: to show endoscopy results at each assessment period.

Analysis item: calculate the number of patients in the analysis groups.

Calculate the number of patients who underwent endoscopy, the number of patients with endoscopy results (normal, remission mucosa, mild, moderate and severe), and the percentage to the patients who underwent endoscopy per assessment period.

Note: Follow "12.3 Assessment period for Mayo score" for Time Allowance of assessment period. The analysis covers only the patients with the assessment applicable to Time Allowance of the first administration and each assessment period.